Page: 1

Protocol Number: CV010010
IND Number: 130,436
EUDRACT Number NA

Date **17-Oct-2016** Revised Date: **06-Sep-2017** 

# Clinical Protocol CV010010

A Study to Assess Safety and Tolerability of Single Oral Doses of BMS-986177 in Patients with ESRD treated with chronic hemodialysis

**Revised Protocol Number: 03** 



This document is the confidential and proprietary information of Bristol-Myers Squibb Company and its global affiliates (BMS). By reviewing this document, you agree to keep it confidential and to use and disclose it solely for the purpose of assessing whether your organization will participate in and/or the performance of the proposed BMS sponsored study. Any permitted disclosures will be made only on a confidential "need to know" basis within your organization or to your independent ethics committee(s). Any other use, copying, disclosure or dissemination of this information is strictly prohibited unless expressly authorized in writing by BMS. Any supplemental information (e.g., amendments) that may be added to this document is also confidential and proprietary to BMS and must be kept in confidence in the same manner as the contents of this document. Any person who receives this document without due authorization from BMS is requested to return it to BMS or promptly destroy it. All other rights reserved. References to BMS in this protocol may apply

| Final Clinical Study Report | CV010010 |
|-----------------------------|---------------|
| MS- 86177 | Factor XIa In |
| Clinical Protocol | CV010010 |
| BMS-986177 | FXIa |

to partners to which BMS has transferred obligations, e.g., a Contract Research Organization (CRO).

Replace all previous version(s) of the protocol with this revised protocol and please provide a copy of this revised protocol to all study personnel under your supervision, and archive the previous versions.

Factor XIa In

Clinical Protocol BMS 986177 CV010010 FXIa

# TABLE OF CONTENTS

| TITLE PAGE | |
|---------------------------------------------------------------|----------|
| DOCUMENT HISTORY | 3 |
| | 4 |
| SUMMARY OF KEY CHANGES FOR REVISED PROTOCOL 03 | 4 |
| TABLE OF CONTENTS | ( |
| 1 SYNOPSIS | 9 |
| 2. SCHEDULE OF ACTIVITIES | 10 |
| 3. INTRODUCTION | 15 |
| | 15 |
| | 16 |
| 3.3 Benefit/Risk Assessment | 17 |
| 4. OBJECTIVES AND ENDPOINTS | 19 |
| 5. STUDY DESIGN | 20 |
| 5.1 Overall Design | 20 |
| 5.1.1 Data Monitoring Committee and Other External Committees | 22 |
| 5.2 Number of Participants | 22 |
| 5.3 End of Study Definition | 22 |
| 5.5 File of Study Definition | 22 |
| | 22 |
| 6. STUDY POPULATION | 24 |
| 6.1 Inclusion Criteria | 24 |
| 6.2 Exclusion Criteria | 25 |
| 6.3 Lifestyle Restrictions | 27 |
| 6.4 Screen Failures | 27 |
| 6.4.1 Retesting During Screening or Lead-In Period | 28 |
| 7. TREATMENT | 28 |
| 7.1 Treatments Administered | 3( |
| | 3( |
| 7.2 Method of Treatment Assignment | 31 |
| 7.3 Blinding | 31 |
| 7.4 Dosage Modification. | 31 |
| 7.5 Preparation/Handling/Storage/Accountability | 31 |
| 7.5.1 Retained Samples for Bioavailability / Bioequivalence | 31 |
| 7.6 Treatment Compliance | 32 |
| 7.7 Concomitant Therapy | |
| 7.7.1 Prohibited and/or Restricted Treatments | 32<br>32 |
| 7.7.2 Other Restrictions and Precautions | |
| 7.8 Treatment After the End of the Study | 32 |
| 8. DISCONTINUATION CRITERIA | 33 |
| 8.1 Discontinuation from Study Treatment | 33 |
| 8.1.1 Post Study Treatment Study Follow-up | 34 |
| 8.2 Discontinuation from the Study | 34 |
| 8.3 Lost to Follow-Up. | 34 |
| 9. STUDY ASSESSMENTS AND PROCEDURES | 35 |
| 9.1 Efficacy Assessments | 35 |

| Clinical Protocol<br>BMS 986177 | CV010010<br>FXIa |
|---|---|
| 9.1.1 Imaging Assessment for the Study. | 35 |
| 9.2 Adverse Events | 35 |
| 9.2.1 Time Period and Frequency for Collecting AE and SAE Information | 35 |
| 9.2.2 Method of Detecting AEs and SAEs | 36 |
| 9.2.3 Follow-up of AEs and SAEs | 36 |
| 9.2.4 Regulatory Reporting Requirements for SAEs | 37 |
| 9.2.5 Pregnancy | 37 |
| 9.2.6 Laboratory Test Result Abnormalities | 37 |
| 9.2.7 Potential Drug Induced Liver Injury (DILI) | 38 |
| 9.2.8 Other Safety Considerations | 38 |
| 9.3 Overdose | 38 |
| 9.4 Safety | 39 |
| 9.4.1 Physical Examinations | 39 |
| 9.4.2 Vital signs | 39 |
| | 39 |
| 9.4.3 Electrocardiograms | 39 |
| 9.4.4 Clinical Safety Laboratory Assessments | 40 |
| 9.4.5 Suicidal Risk Monitoring | 40 |
| 9.4.6 Imaging Safety Assessment | |
| 9.5 Pharmacokinetic | 40 |
| 9.6 Pharmacodynamics | 42 |
| 9.7 Pharmacogenomics | 43 |
| 9.7.1 Genotyping and ADME Sampling | 43 |
| | 43 |
| | 47 |
| | 47 |
| 9.9 Health Economics OR Medical Resource Utilization and Health Economics. | 48 |
| 10. STATISTICAL CONSIDERATIONS | 48 |
| 10.1 Sample Size Determination. | 48 |
| 10.2 Populations for Analyses | 48 |
| 10.3 Statistical Analyses | 48 |
| 10.3.1 Efficacy Analyses | 49 |
| 10.3.2 Safety Analyses | 49 |
| 10.3.3 Pharmacokinetic Analyses | 49 |
| 10.3.4 Other Analyses | 49 |
| 10.3.5 Interim Analyses | 50 |
| 11. REFERENCES | 51 |
| 12 APPENDICES | 53 |
| APPENDIX 1 ABBREVIATIONS AND TRADEMARKS | 54 |
| APPENDIX 2 STUDY GOVERANCE CONSIDERATIONS | 59 |
| APPENDIX 3 ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS: | |
| DEFINITIONS AND PROCEDURES FOR RECORDING, EVALUATING, | |
| FOLLOW UP AND REPORTING. | 67 |
| APPENDIX 4 WOMEN OF CHILDBEARING POTENTIAL DEFINITIONS AND | , |
| METHODS OF CONTRACEPTION | 71 |
| APPENDIX 5 CORE ADME GENE LIST (FROM HTTP://PHARMAADME.ORG) | |
| THE LEVEL SCORE TESTILE GET (FROM THE TIME MANERAL MANERA | 75 |
| | , 5 |
| Revised Protocol No.: 03 | |
| Date: 06 Sep 2017 | 7 |

| Final Clinical Study Report | CV010010 |
|---|---|
| MS- 86177 | Factor XIa In |
| Clinical Protocol<br>BMS 986177 | CV010010<br>FXIa |
| APPENDIX 6 DIAGNOSTIC CRITERIA FOR DRUG<br>APPENDIX 7 REVISED PROTOCOL SUMMARY O | |

| Final Clinical Study Report | CV010010 |
|-----------------------------|---------------|
| MS- 86177 | Factor XIa In |
| Clinical Protocol | CV010010 |
| BMS-986177 | FXIa |

# 1 SYNOPSIS

N/A

# 2. SCHEDULE OF ACTIVITIES

BMS-986177

| Table 21: Proce | dural Outline Sc | reening |
|---|---|---|
| Procedure | Screening<br>Visit (up to 28<br>days prior to<br>First Dose) <sup>a</sup> | Notes |
| Eligibility Assessments | | |
| Informed Consent | x | A participant is considered enrolled only when a protocol specific informed consent is signed. |
| Inclusion/Exclusion Criteria | X | |
| Medical History | x | Include any toxicities or allergy related to previous treatments. |
| Concomitant Medications | X | |
| Safety Assessments | | |
| Physical Examination (PE) | x | If the screening PE is performed within 24 hours prior to dosing on Day 1 then a single exam may count as both the screening and pre-dose evaluation. |
| Physical Measurements | x | Includes height, weight, and BMI. |
| Vital Signs | x | Includes body temperature, respiratory rate, and seated blood pressure and heart rate. Blood pressure and heart rate should be measured after the participant has been resting quietly for at least 5 minutes. |
| Electrocardiogram (ECGs) | х | ECGs should be recorded after the participant has been supine for at least 5 minutes. |
| Laboratory Tests | | |
| Drug Screen (urine or saliva) | x | |
| Alcohol Screen | x | Breathalyzer |
| Clinical Labs | x | Chemistry, CBC, Coagulation and urine dipstick for blood (if participant is able to produce urine). |
| Serology | х | HIV |
| Pregnancy test | x | WOCBP only. See Section 9.4.4. |
| Stool sample for occult blood | x | Subjects may bring sample to the unit on or prior to D1. |
| Adverse Event Reporting | | |
| Monitor for Serious Adverse<br>Events | x | All SAEs must be collected from the date of participant's written consent until 30 days post discontinuation of dosing or participant's participation in the study if the last scheduled visit occurs at a later time. |

a Screening and Day -1 to -3 activities can be combined if performed on the same day

Revised Protocol No.: 03 Date: 06-Sep-2017 FXIa

Clinical Protocol BMS-986177

CV010010 FXIa

**Procedural Outline Treatment** Table 2.-2:

| Procedure | D-1 to-3 | D1 | DS | D8 | D12 | D13 to<br>D15<br>/Study<br>Discharge <sup>a</sup> | Notes |
|---|---|---|---|---|---|---|---|
| Safety Assessments | | | | | | | |
| Physical Examination (PE) | × | | | | | | |
| Targeted PE | | x | × | × | x | X | Targeted physical based on subject complaint. |
| Concomitant Medications | х | х | x | х | x | х | |
| Physical Measurements | × | x | × | × | x | | Weight only. Collect prior to Day 1 visit and collect pre and post dialysis (SoC can be used). |
| Vital Signs | × | × | × | × | × | × | Includes body temperature, respiratory rate, seated blood pressure (BP), and heart rate (HR) on Day-1 to -3 and for those that discontinue prematurely. BP and HR (pre-dose & 3h post HD for all treatments on Days 1, 5, 8, and 12, at 24h post-dose only when BMS-986177 is administered). BP and HR should be measured after the participant has been resting quietly for at least 5 minutes. |
| Electrocardiogram (ECGs) | × | × | × | × | x | | ECGs should be performed prior to Day 1 and conducted 3-6 hours post dialysis. (See note in screening procedures, Section 2) |
| Laboratory Tests | x | x | х | x | x | x | Labs should be obtained prior to Day 1 and obtained 3-6 h post dialysis. (See note in screening procedures, Section 9.4.4.) |
| Stool, occult blood | х | x | x | х | x | | Anytime 2-20 h post-HD. Can bring sample to next HD session. |
| Pregnancy Test | х | | | | | x | WOCBP only. See Section 9.4.4. |
| Urine dipstick | | × | × | × | × | | For blood if urine is produced by the participant. |

Revised Protocol No.: 03 Date: 06-Sep-2017

Ξ

Clinical Protocol BMS-986177

CV010010 FXIa

Procedural Outline Treatment

Table 2.-2:

| Procedure | D-1 to-3 | D1 | DS | 80 | D12 | D13 to<br>D15<br>/Study | Notes |
|---|---|---|---|---|---|---|---|
| | | | | | | Discharge <sup>a</sup> | |
| | | | | | | | Obtain Pre-dose if possible; anytime up to 2-20 h post HD if possible. |
| Drug Test (urine or saliva or plasma) | × | | | | | | |
| Alcohol screen | | x | x | x | x | | Breathalyzer; Pre-dose |
| Adverse Event Reporting | | | | | | | |
| Monitor for Non-Serious<br>Adverse Events | | x | x | x | x | х | AE collection to begin 3 hours prior to dialysis start on Day 1 regardless of study drug administered |
| Monitor for Serious Adverse<br>Events | x | x | x | x | x | х | See note in screening procedures. |
| Pharmacokinetic (PK) Assessments | | | | | | | |
| Serial Blood PK Sampling | | x | x | х | х | | See Section 9.5. PK only being collected on days |
| Single PK Sampling | | | Obtained 2 | Obtained 24-72 hours after each dose | after each d | eso | when BMS-986177 is administered depending on randomization. |
| Pharmacodynamic (PD)<br>Assessments | | | | | | | |
| Serial Blood PD Sampling | | x | x | x | x | | See Section 9.6 and Table 9.6-1 (for BMS-986177 and enoxaparin) and Table 9.6-2 (for UFH). |
| Single PD Sampling | | Obtained | d 24-72 ho | Obtained 24-72 hours after each dose of BMS-986177 only. | h dose of B | MS-986177 | Only after BMS-986177 dosing. See Section 9.6 and Table 9.6-1. |
| Biomarker Assessments | | | | | | | |
| D-dimer, F1,2 and exploratory plasma sample | | x | x | x | × | | See Section 9.8 and Table 9.8-1 and Table 9.8-2. |


12

Factor XIa Inhibitor

CV010010 FXIa

Clinical Protocol BMS-986177

**Procedural Outline Treatment** Table 2.-2:

| Procedure | D-1 to-3 | D 1 | DS | 8Q | D12 | D13 to<br>D15<br>/Study<br>Discharge <sup>a</sup> | Notes |
|---|---|---|---|---|---|---|---|
| FXI antigen | | x | | | | | See Section 9.8 and Table 9.8-1 and Table 9.8-2. |
| Clotting assessment for dialysis filter, drip chamber; dialysis circuit pressure; number and volume of saline flushes; Kt/V, Time to hemostasis at puncture site | | × | × | × | × | | See Section 9.8 and Table 9.8-1 and Table 9.8-2. Clotting Assessment to be conducted by a blinded staff member. |
| Retain dialysis filter | | x | × | х | x | | See Section 9.8. |
| Whole Blood Collection for<br>Analysis of DNA Variants in<br>ADME-related Genes and<br>thrombosis and hemostasis<br>related genes | x | | | | | | See Section 9.7. Only one sample required per subject for the study. Maybe obtained any time on or after randomization |
| Additional Research<br>Sampling | | x | x | x | x (24-72<br>L | x (24-72 h post dose<br>D12) | Residual samples from biomarkers and PD blood. See Section 9.8.1. |
| Clinical Drug Supplies | | | | | | | |
| Randomize | × | | | | | | Visit can be conducted with scheduled HD session. |
| Study Drug Administration | | × | × | x | x | | Administration of study drugs (i.e., BMS-986177, enoxaparin, and UFH) will be depending on the randomized sequence the subject is assigned to. |

<sup>&</sup>lt;sup>a</sup> Visit can be performed between D13-15 based on last PK sample obtained between 24-72 hours post D12 dose. End of study procedures should be performed for subjects that discontinue prematurely.

In the event of multiple procedures are required at a single time point, the following is a list of procedures from highest priority to


13

| CV010010 | Factor XIa Inhibitor |
|-----------------------------|----------------------|
| | 1 |
| Final Clinical Study Report | BMS-986177 |

| CV010010<br>FXIa | | 41 |
|---|---|---|
| | ag<br>ling | |
| | tic Samplii<br>amic Samp<br>npling | : 03 |
| Clinical Protocol<br>BMS-986177 | Safety Pharmacokinetic Sampling Pharmacodynamic Sampling Biomarker sampling | Revised Protocol No.: 03<br>Date: 06-Sep-2017 |
| Clinical Protoc<br>BMS-986177 | Saf Pha Pha Pha Bio | Revised<br>Date: 06 |

Clinical Protocol
BMS-986177
CV010010
FXIa



# 3.1 Study Rationale

Patients with end-stage renal disease (ESRD) in chronic treatment with hemodialysis (HD), are administered anticoagulant agents before and during the HD sessions to prevent clotting of the extracorporeal circuit. Clot formation in the hemodialysis circuit can reduce the efficiency of the procedure and, in the most severe cases, lead to complete occlusion of the lines or the hemodialytic filter with the consequent interruption of the HD and blood loss for the patient. Guidelines for clotting prevention recommend unfractionated heparin (UFH) or low-molecular-

weight heparin such as enoxaparin, is administered during the HD session. However, UFH and LMWH can potentially increase the hemorrhagic risk in patients with ESRD who frequently exhibit a uraemia-associated platelet dysfunction. Furthermore, some patients treated with heparins develop anti-heparin antibodies causing an autoimmune disorder called heparin-induced thrombocytopenia (HIT) that prevents further use of heparin. In this regard, FXIa inhibition might represent an alternative and safer anticoagulant option in patients undergoing HD in whom heparin administration is not indicated. Anti-coagulant agents are utilized in clinical practice to reduce the incidence of thrombotic agents in several conditions, and although effective in preventing thrombus formation, they are also associated with dose-related bleeding complications. Observations from patients with genetic deficit of FXI and from clinical and preclinical studies that investigated this mechanism of action suggest that inhibition of FXIa may be safer in terms of bleeding risk compared to other anti-coagulants. If this is confirmed, BMS-986177 may in the future be also used to prevent or treat thrombotic events. Thus, this study will also provide relevant information on the anticoagulant activity of BMS-986177 compared to two different comparators (UFH and enoxaparin) that are routinely used in several thrombotic conditions.

## Research hypothesis

The purpose of this study is to evaluate the safety profile, tolerability, and pharmacokinetics of single oral doses of BMS-986177 in ESRD patients undergoing chronic stable hemodialysis treatment. Although there is no primary research hypothesis to be formally tested, it is expected that administration of BMS-986177 will prolong the plasma activated partial thromboplastin time (aPTT), reduce plasma Factor XI clotting activity, and have no effect on the prothrombin time and international normalized ratio (PT and INR).

It is expected that the administration of BMS-986177 will prevent clot formation in the extracorporeal HD circuit, hence clotting in the HD filter, lines, and drip chambers will be assessed, additional clotting-related pharmacodynamic (PD) endpoints will be also explored.



clinically apparent bleeding or bruising; puncture sites will be closely monitored and patients will be discharged from the study unit only once hemostasis at those sites has been reached. Additionally, phlebotomy may cause blood clots, discomfort, and/or inflammation at the respective sites.

Patients' progression in the study will depend on the clinical safety profile, including reported AEs, findings from physical examinations, clinical laboratory results, vital signs, and ECGs of all previous arms to and including the preceding dose.

A study of pharmacokinetic of BMS-986177 in patients with severe renal impairment undergoing hemodialysis (CV010-012) is ongoing. Data from the first 4 patients of CV010-012 have been analyzed to characterize PK and dialytic clearance in this patient population. The results from this modeling and simulation guided final dose selection for this study to attain target concentrations and avoid exceeding target exposures (see Section 5.5 Justification for Dose).

Reproductive toxicology studies have been performed for BMS-986177 and support, women of child-bearing potential (WOCBP) to be included in the study (For additional information refer to the Investigator's Brochure). WOCBP undergoing dialysis receive UFH or LMWH. All WOCBP will be monitored for pregnancy.

In summary, the overall safety profile of BMS-986177 in non-clinical and clinical studies supports further evaluation of the safety, tolerability, PK profile, and pharmacodynamic (PD) responses in ESRD patients undergoing HD. While the adverse effects observed in nonclinical studies at high multiple of exposure were not observed in healthy volunteers, these signals (LFTs) will be monitored in the setting of the current clinical study. All patients will be informed of the potential risks prior to enrollment in the study

# 4. OBJECTIVES AND ENDPOINTS

Table 4.-1: Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| <ul> <li>To assess safety and tolerability of single oral doses of BMS-986177 in<br/>patients with end-stage renal disease on chronic hemodialysis treatment.</li> </ul> | AEs, clinical laboratory<br>values, vital signs, ECGs. |
| Secondary | |
| <ul> <li>To characterize the pharmacokinetic profile of BMS-986177 in a<br/>hemodialysis population, and determine the extent of BMS-986177 on<br/>dialytic removal.</li> </ul> | Cmax, AUC, dialytic clearance. |

Protocol No.: 03 Date: 06-Sep-2017

Table 4.-1: Objectives and Endpoints

| Objectives | End | lpoints |
|------------|-----|---------|

### STUDY DESIGN

# 5.1 Overall Design

This study is a multicenter, cross-over, randomized, open-label trial with blinded endpoint assessment investigating safety and tolerability of single oral doses of BMS-986177 in patients with ESRD undergoing chronic stable HD three times per week. Secondary objectives are to assess BMS-986177 pharmacokinetics and hemodialysis success defined as completion of hemodialysis without premature interruption of the procedure due to complete clotting of the dialytic circuit and/or filter.

Study treatments will be administered on the first and last HD day of the week (either Monday and Friday, or Tuesday and Saturday, depending on the patients HD schedule), for a total of 4 treatment days (2 doses of BMS-986177, 1 dose of UFH, 1 dose of Enoxaparin).

The 2nd HD day of the week is not a study treatment day; on that day, study patients will undergo dialysis with standard of care, as per their schedule, and no study activities will be performed on those days.

Screening for inclusion in the study will be performed up to 28 days before the first study visit. After screening and meeting eligibility as per inclusion and exclusion criteria, patients will be randomized to 1 of following 4 sequences that will be conducted in parallel.

| Sequence No. | Period | | | |
|--------------|-------------|-------------|-------------|-------------|
| | 1 | 2 | 3 | 4 |
| 1 | UFH | BMS dose 1 | BMS dose 2 | Enoxaparin |
| | | (BMS-986177 | (BMS-986177 | |
| | | 100 mg) | 300 mg) | |
| 2 | BMS dose 1 | Enoxaparin | UFH | BMS dose 2 |
| | (BMS-986177 | | | (BMS-986177 |
| | 100 mg) | | | 300 mg) |
| 3 | BMS dose 2 | UFH | Enoxaparin | BMS dose 1 |
| | (BMS-986177 | | | (BMS-986177 |
| | 300 mg) | | | 100 mg) |
| 4 | Enoxaparin | BMS dose 2 | BMS dose 1 | UFH |
| | | (BMS-986177 | (BMS-986177 | |
| | | 300 mg) | 100 mg) | |

Note: Per amendment/revised protocol 01, the BMS-986177 doses will be 100 mg (BMS dose 1) and 300 mg (BMS dose 2).

Study patients will be admitted to the study facility the same day of HD treatment day or the night before. Assessment of vital signs and clinical biochemistry will be performed pre-dose.

Study treatments will be administered:

- BMS-986177: one single oral dose 3 hours prior beginning the HD session
- UFH: I.V. infusion to start within 10 minutes prior beginning the HD session. The dosage and duration of UFH use are at the discretion of the physicians and are per their institutional practice.
- Enoxaparin: one single dose (40 mg) by subcutaneous injection 3 hours prior beginning the HD session

The HD session will last approximately 4 hours. However, the duration could range from 3 to 4 hours but should be consistent on the days when study drug is administered. After the HD, patients will remain in the study facility for at least:

- Approximately 3 hours post-HD on UFH and Enoxaparin treatment days
- Approximately 24 hours post-dose on BMS-986177 days

Site staff members blinded to treatment will perform an assessment of clot formation according to criteria set forth in the Clot Formation Assessment Manual which will be provided to the site in a separate document.

Physical examinations, vital sign measurements, 12-lead electrocardiograms (ECG), and clinical laboratory evaluations will be performed at selected times throughout the dosing interval. Participants will be closely monitored for adverse events throughout the study. Blood samples will be collected for up to 72 hours after study drug administration for pharmacokinetic (PK) analysis and pharmacodynamic (PD) analysis. Approximately 365 mL of blood will be drawn from each participant during the study.

The study design schematic is presented in Figure 5.1-1.

**Figure 5.1-1:** Study Design Schematic

| | | Week 1 | | | | | | Week 2 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | D-21 to D-1 | D1* | D2 | D3 | D4 | D5‡ | D6 | D7 | D8* | D9 | D10 | D11 | D12‡ | D13 to D15 |
| HD<br>days | | 1 <sup>st</sup><br>HD | | 2 <sup>nd</sup><br>HD | | 3 <sup>rd</sup><br>HD | | | 1 <sup>st</sup><br>HD | | 2 <sup>nd</sup><br>HD | | 3 <sup>rd</sup><br>HD | |
| Study activity | S-E-R | Tx | | | | Tx | | | Tx | | | | Tx | D |

HD = Hemodialysis session. S= Screening. E = Enrollment. R = Randomization. Tx = Study treatment day (BMS-986177 dose 1 or dose 2, or unfractionated heparin, or enoxaparin). D = Study discharge.


**FXIa** 

<sup>\*</sup> D1 and D8 can be Monday or Tuesday depending on the patient's dialysis schedule.

<sup>&</sup>lt;sup>‡</sup>D5 and D12 can be Friday or Saturday depending on the patient's dialysis schedule.

Note: Per amendment/revised protocol 01, the BMS-986177 doses will be 100 mg (BMS dose 1) and 300 mg (BMS dose 2).

# 5.1.1 Data Monitoring Committee and Other External Committees

Not Applicable

# 5.2 Number of Participants

Target sample size is 32 participants to achieve 24 participants who completed the 4 study treatments.

# 5.3 End of Study Definition

The start of the trial is defined as the first visit for first participant screened. End of trial is defined as the last visit or scheduled procedure shown in the Schedule of Activities for the last participant. Study completion is defined as the final date on which data for the primary endpoint was or is expected to be collected.



Final Clinical Study Report CV010010
BMS-986177 Factor XIa Inhibitor

Clinical Protocol CV010010
BMS-986177 FXIa



## 6. STUDY POPULATION

For entry into the study, the following criteria MUST be met.

# 6.1 Inclusion Criteria

## 1) Signed Written Informed Consent

a) The signed informed consent form.

# 2) Type of Participant and Target Disease Characteristics

- a) Subjects with ESRD treated with hemodialysis prescribed 3 times a week for at least 3 months prior enrollment. For at least 2 weeks prior to study drug administration, participants should undergo all 3 hemodialysis sessions per week.
- b) Subjects with severe renal impairment may include those with a variety of underlying stable renal disease such as nephrosclerosis and chronic glomerulonephritis.

### 3) Age and Reproductive Status

- a) Males and Females, ages 18 or age of majority to 75 years, inclusive
- b) Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
- c) Women must not be breastfeeding
- d) Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception (Appendix 4) for the duration of the study plus 5 half-lives of study treatment BMS-986177 (2 days) plus 30 days (duration of ovulatory cycle) for a total of 32 days post-treatment completion.
- e) Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (Appendix 4) for the duration of treatment with study treatment(s) BMS-986177 plus 5 half-lives of the study treatment (2 days) plus 90 days (duration of sperm turnover) for a total of 92 days post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.
  - i) With amendment/revised protocol 02, males who are sexually active with WOCBP must agree to follow instructions for methods of contraception (Appendix 4) for the duration of treatment with BMS-996177 plus 5 half-lives of the study treatment (2 days) for a total of 2 days post-treatment completion.
- f) Azoospermic males are exempt from contraceptive requirements. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, and still must undergo pregnancy testing as described in this section.

Investigators shall counsel WOCBP, and male participants who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception, (Appendix 4) which have a failure rate of < 1% when used consistently and correctly.

#### 6.2 Exclusion Criteria

#### 1) Medical Conditions

- a) Subjects receiving dialysis through central venous catheters. After amendment/revised protocol 01, this exclusion criteria will not be applicable and will not be needed for eligibility.
- b) History of uncontrolled or unstable cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematopoietic, psychiatric and/or neurological disease in the past 3 months
- c) Evidence or history of coagulopathy, prolonged or unexplained clinically significant bleeding, or frequent unexplained bruising.
- d) Current or recent (within 3 months of study drug administration) gastrointestinal disease or surgery, which by the judgment of the Investigator, may increase a subject's risk of gastrointestinal bleeding or interfere with absorption of study drug (eg, peptic or gastric ulcer disease, severe gastritis, history of gastrointestinal surgery with the exception of history of cholecystectomy).


Clinical Protocol BMS-986177 CV010010 FXIa

- e) Any condition requiring chronic systemic anticoagulation such as, but not limited to, atrial fibrillation, mechanical prosthetic valve, deep venous thrombosis, or pulmonary embolism
- f) Not considered by the study principal investigator to be candidates for oral anticoagulation (for example, history of intracranial hemorrhage, active bleeding, recent gastrointestinal bleed or retroperitoneal bleed, severe hepatic impairment)
- g) Any major surgery within 12 weeks of study drug administration
- h) History of significant head injury within the last 2 years, including subjects with base of skull fractures
- i) Donation of blood to a blood bank within 4 weeks of study drug administration (within 2 weeks for plasma only)
- j) Blood transfusion within 2 weeks of study drug administration
- k) Inability to tolerate oral medication
- 1) Inability to be venipunctured and/or tolerate venous access
- m) Smoking more than 10 cigarettes per day
- n) Recent (within 6 months of study drug administration) drug or alcohol abuse as defined in DSM IV, Diagnostic Criteria for Drug and Alcohol Abuse (Appendix 6)
- o) Any other sound medical, psychiatric and/or social reason as determined by the investigator

### 2) Prior/Concomitant Therapy

- a) Chronic therapy with aspirin, dipyridamole, or P2Y12 antagonists (for example clopidogrel, prasugrel, or ticagrelor). Prior aspirin use is allowed after a washout period of at least 1 week before dosing.
- b) Inability to comply with prohibited/restricted treatments as listed in Section 7.7

#### 3) Physical and Laboratory Test Findings

- a) Evidence of organ dysfunction or any clinically significant deviation in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with their degree of renal dysfunction and other underlying conditions as determined by medical history, physical examination, ECG, and clinical laboratory determinations.
- b) Subjects with macro-hematuria and/or fecal occult blood detected during screening, baseline, or documented during other recent medical assessment, unless deemed not clinically significant by the Investigator.
- c) Subjects at screening with the following abnormal laboratory values upon repeat testing are excluded:
  - i) Hemoglobin <9 g/dL
  - ii) Hematocrit < 30%
  - iii) Platelet count < 80,000/mm<sup>3</sup>
  - iv) ALT or AST > ULN
  - v) Total bilirubin > 1.5X ULN
  - vi) aPTT or PT/INR > 1.2X ULN

- d) Positive urine or saliva or plasma screen for drugs of abuse with exception for prescription medications
- e) Positive blood screen for HIV-1 and HIV-2 antibody

### 4) Allergies and Adverse Drug Reaction

a) History of any significant drug allergy (such as anaphylaxis or hepatotoxicity)

### 5) Other Exclusion Criteria

- a) Prisoners or participants who are involuntarily incarcerated. (Note: under certain specific circumstances a person who has been imprisoned may be included or permitted to continue as a participant. Strict conditions apply and Bristol-Myers Squibb approval is required.)
- b) Participants who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Eligibility criteria for this study have been carefully considered to ensure the safety of the study participants and that the results of the study can be used. It is imperative that participants fully meet all eligibility criteria.

### 6.3 Lifestyle Restrictions

Subjects are to refrain from strenuous exercise, contact sports, and sunbathing from at least 5 day(s) prior to the first dose until study discharge.

- 1) Unless restricted by the clinical facility, subjects are permitted to smoke while residing at the clinical facility and on dialysis days.
- 2) Participants are not permitted to consume alcohol-containing beverages from 3 days prior to the first dose until study discharge.
- 3) Participants are not permitted to consume grapefruit-containing products from 3 days prior to the first dose until study discharge.
- 4) Participants are not permitted to consume more than two caffeine-containing beverages per day for the whole study duration.
- 5) On each study treatment day, patients are required to fast (nothing to eat or drink except water) for 4 hours prior to a standard meal, which will be consumed approximately 30 minutes prior to study drug administration. Patients may not drink water one hour before and after study drug administration except with dosing and the beverage provided with the pre-dose standard meal. Water may be consumed *ad libitum* at other times.

#### 6.4 Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently [randomized/entered in the study/included in the analysis population]. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants, to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements, and to respond to queries from regulatory authorities. Minimal

information includes date of consent, demography, screen failure details, eligibility criteria, and any serious AEs.

# 6.4.1 Retesting During Screening or Lead-In Period

Participant Re-enrollment: This study permits the re-enrollment of a participant that has discontinued the study as a pre-treatment failure (i.e., participant has not been randomized / has not been treated). If re-enrolled, the participant must be re-consented.

Laboratory parameters and/or assessments that are included in Table 2.-1, Screening Procedural Outline may be repeated in an effort to find all possible well-qualified participants. Consultation with the Medical Monitor may be needed to identify whether repeat testing of any particular parameter is clinically relevant.

#### 7. TREATMENT

Study treatment is defined as any investigational treatment(s), marketed product(s), placebo or medical device intended to be administered to a study participant according to the study randomization or treatment allocation.

Study treatment includes both Investigational [Medicinal] Product (IP/IMP) and Non-investigational [Medicinal] Product (Non-IP/Non-IMP) and can consist of the following:

BMS-986177, unfractionated heparin (UFH) and Enoxaparin as IP/IMP.

An investigational product, also known as investigational medicinal product in some regions, is defined a pharmaceutical form of an active substance or placebo being tested or used as a reference in a clinical study, including products already with a marketing authorization but used or assembled (formulated or packaged) differently than the authorized form, or used for an unauthorized indication, or when used to gain further information about the authorized form.

Other medications used as support or escape medication for preventative, diagnostic, or therapeutic reasons, as components of the standard of care for a given diagnosis, may be considered as non-investigational products. Not Applicable for this study.

Factor XIa Inhibitor

Clinical Protocol BMS-986177

CV010010 FXIa

Study treatments for CV010010

**Table 7.-1:** 

| roduct Description /<br>Class and Dosage<br>Form | Potency | dMI-noN/dI | Blinded or Open<br>Label | Packaging /<br>Appearance | Storage Conditions<br>(per label) |
|---|---|---|---|---|---|
| SMS 986177/SDD<br>75% as the base <sup>a</sup> | 100 mg or 300 mg | ď | Open label | Labeled bulk product in glass vials / white to off-white powder which may appear as lumps | Store at 2 C to 8 C, protected from light and moisture |
| UFH | Per Standard of Care | Ш | Open label | Sourced by Site | PerLabel |
| Enoxaparin | 40 mg | II. | Open label | Sourced by Site | Per Label |

<sup>&</sup>lt;sup>a</sup> Compounding instructions will be provided separately to the site

59

601

### 7.1 Treatments Administered

Table 7.1-1: Selection and Timing of Dose

| Study Treatment | Unit dose<br>strength(s)/Dosage<br>level(s) | Dosage formulation<br>Frequency of<br>Administration | Route of Administration |
|---|---|---|---|
| Dose 1<br>BMS 986177/SDD<br>75% as the base <sup>a</sup> | 100 mg | Single dose | РО |
| Dose 2<br>BMS 986177/SDD<br>75% as the base <sup>a</sup> | 300 mg | Single dose | РО |
| UFH | Per SoC | (Standard of Care) | IV |
| Enoxaparin | 40 mg | Single Dose<br>(Standard of Care) | SC |

a Compounding instructions will be provided separately to the site

Note: Per amendment/revised protocol 01, the BMS-986177 doses will be 100 mg (BMS dose 1) and 300 mg (BMS dose 2).

Study treatments will be dosed:

- BMS-986177: one single oral dose 3 hours prior beginning the HD session
- UFH: I.V. infusion to start within 10 minutes prior beginning the HD session. The dosage and duration of UFH use are at the discretion of the physicians and are per their institutional practice.
- Enoxaparin: one single dose (40 mg) by subcutaneous injection 3 hours prior beginning the HD session

At the time of dosing, BMS-986177, 240 mL of water will be administered to the participant along with his/her dose of study drug. The time of dose administration will be called "0" hour.

Restrictions related to food and fluid intake are described in Section 6.3.

# 7.2 Method of Treatment Assignment

Study treatment will be dispensed at the study visits as listed in Schedule of Activities (Section 2).

Enrolled participants, including those not dosed, will be assigned sequential participant numbers starting with 00001, (eg, 00001, 00002, 00003.... 00010). Sequential numbering may restart at 00001 for each participating site as the distinct patient identification number (PID) will ultimately be comprised of the site number and participant number, (eg, 0002 00001). Those enrolled participants meeting inclusion and exclusion criteria will be eligible to be randomized. Randomization numbers will be assigned prior to dosing.

Participants will not be replaced if they are discontinued from the study secondary to an adverse event unless the adverse event can be determined to be unrelated to treatment. If a participant is replaced after dosing then the replacement participant will be assigned the original participant's number plus 100. The replacement participant will receive the same treatment as the participant being replaced but a new randomization number will be assigned to him or her. For example, participant 4 would be replaced by Participant 104.

# 7.3 Blinding

This is an open-label study. Blinding procedures are not applicable.

# 7.4 Dosage Modification

Not Applicable

## 7.5 Preparation/Handling/Storage/Accountability

The investigational product should be stored in a secure area according to local regulations. It is the responsibility of the investigator to ensure that investigational product is only dispensed to study Participants. The investigational product must be dispensed only from official study sites by authorized personnel according to local regulations.

The product storage manager should ensure that the study treatment is stored in accordance with the environmental conditions (temperature, light, and humidity) as determined by BMS. If concerns regarding the quality or appearance of the study treatment arise, the study treatment should not be dispensed and contact BMS immediately.

Study treatment not supplied by BMS will be stored in accordance with the package insert.

Investigational product documentation (whether supplied by BMS or not) must be maintained that includes all processes required to ensure drug is accurately administered. This includes documentation of drug storage, administration and, as applicable, storage temperatures, reconstitution, and use of required processes (eg, required diluents, administration sets).

For study drugs not provided by BMS (enoxaparin and UFH) and obtained commercially by the site, storage should in accordance with the product label.

Compounding instructions for BMS-986177 will be provided separately to the site.

 Further guidance and information for final disposition of unused study treatment are provided in Appendix 2.

#### 7.5.1 Retained Samples for Bioavailability / Bioequivalence

Not Applicable

# 7.6 Treatment Compliance

Study drug will be administered in the clinical facility. After administration of BMS-986177 an examination of the oral cavity is required to verify that a participant has swallowed the solution. The participant should drink the entire aliquot of water given to swallow the solution.

UFH and Enoxaparin will be administered by the healthcare staff at the clinical facility according to protocol and standard of care.

# 7.7 Concomitant Therapy

#### 7.7.1 Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications taken prior to study drug administration in the study are described below. Medications taken within 4 weeks prior to study drug administration must be recorded on the CRF.

- 1) Use of any agent, including but not limited to anti-platelet agents (except aspirin), anticoagulants (except heparin for routine hemodialysis use), fish oil capsules, and ginko that is known to increase the potential for bleeding within 2 weeks prior to study drug administration. Use of non-steroidal anti-inflammatory compounds (NSAIDs) or aspirin within 1 week prior to study drug administration.
- 2) Exposure to any investigational drug or placebo within 4 weeks of study drug administration.
- 3) Use of acid controllers within two days of BMS-986177 study drug administration except those medications cleared by the BMS medical monitor. The use of acid controllers after BMS-986177 administration and after hemodialysis is allowed. The use of acid controllers is also allowed when enoxaparin or UFH are administered.
  - a) Sodium bicarbonate is allowed during the study.
- 4) Use of strong and moderate CYP3A inhibitors within 1 week of enrollment including the following: the antifungals and antibiotics ketoconazole, fluconazole, itraconazole, miconazole, clotrimazole, erythromycin and clarithromycin; the calcium channel blockers diltiazem and verapamil; the HIV anti-virals delaviridine, indinavir, nelfinavir, ritonavir, and saquinavir; and the serotonin reuptake inhibitor fluoxetine. Use of CYP3A inducers such as carbamazapine, dexamethasone, phenobarbitol, phenytoin, rifampin, St John's Wort within 4 weeks of enrollment. Topical antifungal use is allowed.

Study patients may receive treatment with medications necessary for maintaining the clinical status of their condition as described in Inclusion Criteria.

Any concomitant therapies must be recorded on the CRF.

#### 7.7.2 Other Restrictions and Precautions

Not Applicable

#### 7.8 Treatment After the End of the Study

At the end of the study, BMS will not continue to provide BMS supplied study treatment to participants/investigators unless BMS chooses to extend the study. The investigator should ensure that the participant receives appropriate standard of care to treat the condition under study.

#### 8. DISCONTINUATION CRITERIA

# 8.1 Discontinuation from Study Treatment

Participants MUST discontinue investigational product (and non-investigational product at the discretion of the investigator) for any of the following reasons:

- Participant's request to stop study treatment. Participants who request to discontinue study
  treatment will remain in the study and must continue to be followed for protocol specified
  follow-up procedures. The only exception to this is when a participant specifically withdraws
  consent for any further contact with him/her or persons previously authorized by participant
  to provide this information
- Any clinical adverse event (AE), laboratory abnormality or intercurrent illness which, in the
  opinion of the investigator, indicates that continued participation in the study is not in the
  best interest of the participant
- Termination of the study by Bristol-Myers Squibb (BMS)
- Loss of ability to freely provide consent through imprisonment or involuntarily incarceration for treatment of either a psychiatric or physical (eg, infectious disease) illness
- Pregnancy
- Overt bleeding producing a Hb decrease ≥ 2 g/dL in 24 hours
- Need for blood transfusion
- Overt bleeding which is retroperitoneal, intracranial, intra-spinal, intraocular, or intraarticular
- Any overt bleeding deemed by the investigator to necessitate discontinuation of trial medication
- Medical or surgical treatment for bleeding beyond the application of pressure or cold compress
- Need for surgery during the study period
- Need for treatment with an anticoagulant or antiplatelet agent during the study period, with the exception of heparin and enoxaparin use during HD
- Need for treatment with a strong CYP3A4 inhibitor or any CYP3A4 inducers
- Inability to continue on the hemodialysis treatment for the duration of the study
- Inability to comply with the protocol
- Occurrence in one of the BMS-986177 treatment arm or in the enoxaparin treatment arm of 5 or more patients with events of complete clotting of HD circuit causing premature interruption of the HD procedure. This will result in a discontinuation of that treatment arm. The randomized sequence for the following patients will not be changed, and the discontinued treatment arm will be replaced by standard of care (UFH) in the treatment sequence.

In case a subject experiences complete clotting leading to premature interruption of HD in the BMS-986177 arms, the HD session can be restarted using standard of care at the discretion of the study Investigator.

Refer to the Schedule of Activities for data to be collected at the time of treatment discontinuation and follow-up and for any further evaluations that can be completed

All participants who discontinue study treatment should comply with protocol specified follow-up procedures as outlined in Section 2. The only exception to this requirement is when a participant withdraws consent for all study procedures including post-treatment study follow-up or loses the ability to consent freely (i.e., is imprisoned or involuntarily incarcerated for the treatment of either a psychiatric or physical illness).

If study treatment is discontinued prior to the participant's completion of the study, the reason for the discontinuation must be documented in the participant's medical records and entered on the appropriate case report form (CRF) page.

## 8.1.1 Post Study Treatment Study Follow-up

Participants who discontinue study treatment may continue to be followed.

## 8.2 Discontinuation from the Study

Participants who request to discontinue study treatment will remain in the study and must continue to be followed for protocol specified follow-up procedures. The only exception to this is when a participant specifically withdraws consent for any further contact with him/her or persons previously authorized by participant to provide this information.

- Participants should notify the investigator of the decision to withdraw consent from future follow-up in writing, whenever possible.
- The withdrawal of consent should be explained in detail in the medical records by the
  investigator, as to whether the withdrawal is from further treatment with study treatment only
  or also from study procedures and/or post treatment study follow-up, and entered on the
  appropriate CRF page.
- In the event that vital status (whether the participant is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.
- If the participant withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such a withdrawal of consent.

#### 8.3 Lost to Follow-Up

- All reasonable efforts must be made to locate participants to determine and report their ongoing status. This includes follow-up with persons authorized by the participant.
- Lost to follow-up is defined by the inability to reach the participant after a minimum of three
  documented phone calls, faxes, or emails as well as lack of response by participant to one
  registered mail letter. All attempts should be documented in the participant's medical
  records.
- If it is determined that the participant has died, the site will use permissible local methods to obtain date and cause of death.
- If investigator's use of third-party representative to assist in the follow-up portion of the study has been included in the participant's informed consent, then the investigator may use a Sponsor retained third-party representative to assist site staff with obtaining participant's contact information or other public vital status data necessary to complete the follow-up portion of the study.

- The site staff and representative will consult publicly available sources, such as public health registries and databases, in order to obtain updated contact information.
- If after all attempts, the participant remains lost to follow-up, then the last known alive date
  as determined by the investigator should be reported and documented in the participant's
  medical records.

#### 9. STUDY ASSESSMENTS AND PROCEDURES

- Study procedures and timing are summarized in the Schedule of Activities.
- Protocol waivers or exemptions are not allowed.
- All immediate safety concerns must be discussed with the Sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue treatment.
- Adherence to the study design requirements, including those specified in the Schedule of Activities, is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential
  participants meet all eligibility criteria before randomization. The investigator will maintain a
  screening log to record details of all participants screened and to confirm eligibility or record
  reasons for screening failure, as applicable.
- Procedures conducted as part of the participant's routine clinical management (eg, blood count) and obtained before signing of informed consent may be utilized for screening or baseline purposes provided the procedure meets the protocol-defined criteria and has been performed within the timeframe defined in the Schedule of Activities.

## 9.1 Efficacy Assessments

Not Applicable

### 9.1.1 Imaging Assessment for the Study

Not Applicable

### 9.2 Adverse Events

The definitions of an AE or serious adverse event (SAE) can be found in Appendix 3.

AEs will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).

The investigator and any designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study treatment or the study, or that caused the participant to discontinue before completing the study.

#### SAE reporting specified in Appendix 3

# 9.2.1 Time Period and Frequency for Collecting AE and SAE Information

The collection of nonserious AE information should begin at initiation of study treatment until [the follow-up contact], at the timepoints specified in the Schedule of Activities (Section 2).

Nonserious AE information should also be collected from the start of a placebo lead-in period or other observational period intended to establish a baseline status for the participants.

Sections 5.6.1 and 5.6.2 in the Investigator Brochure (IB) represent the Reference Safety Information to determine expectedness of serious adverse events for expedited reporting. Following the participant's written consent to participate in the study, all SAEs, whether related or not related to study drug, must be collected, including those thought to be associated with protocol-specified procedures.

All SAEs must be collected that occur during the screening period and within 30 days of discontinuation of dosing.

- Medical occurrences that begin before the start of study treatment but after obtaining informed consent will be recorded on the appropriate section of the eCRF section.
- All SAEs will be recorded and reported to Sponsor or designee within 24 hours, as indicated in Appendix 3.
- The investigator will submit any updated SAE data to the sponsor within 24 hours of this being available.

Investigators are not obligated to actively seek AEs or SAEs in former study participants. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event reasonably related to the study treatment or study participation, the investigator must promptly notify the sponsor.

The method of evaluating, and assessing causality of AEs and SAEs and the procedures for completing and reporting/transmitting SAE reports are provided in Appendix 3.

# 9.2.2 Method of Detecting AEs and SAEs

Adverse events can be spontaneously reported or elicited during open-ended questioning, examination, or evaluation of a subject. (In order to prevent reporting bias, subjects should not be questioned regarding the specific occurrence of one or more AEs.)

### 9.2.3 Follow-up of AEs and SAEs

- Nonserious AEs should be followed to resolution or stabilization, or reported as SAEs if they become serious (see Appendix 3).
- Follow-up is also required for nonserious AEs that cause interruption or discontinuation of study treatment and for those present at the end of study treatment as appropriate.
- All identified nonserious AEs must be recorded and described on the nonserious AE page of the CRF (paper or electronic). Completion of supplemental CRFs may be requested for AEs and/or laboratory abnormalities that are reported/identified during the course of the study.

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All SAEs, and non-serious AEs of special interest (as defined in Section 9.2 will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the participant is lost to follow-up (as defined in Section 8.3).
Further information on follow-up procedures is given in Appendix 3.

# 9.2.4 Regulatory Reporting Requirements for SAEs

- Prompt notification by the investigator to the Sponsor of SAEs is essential so that legal
  obligations and ethical responsibilities towards the safety of participants and the safety of a
  product under clinical investigation are met.
- An investigator who receives an investigator safety report describing SAEs or other specific safety information (e.g., summary or listing of SAEs) from the Sponsor will file it along with the Investigator's Brochure and will notify the IRB/IEC, if appropriate according to local requirements.

Sponsor or designee will be reporting adverse events to regulatory authorities and ethics committees according to local applicable laws including European Directive 2001/20/EC and FDA Code of Federal Regulations 21 CFR Parts 312 and 320. A SUSAR (Suspected, Unexpected Serious Adverse Reaction) is a subset of SAEs and will be reported to the appropriate regulatory authorities and investigators following local and global guidelines and requirements.

# 9.2.5 Pregnancy

If, following initiation of the study treatment, it is subsequently discovered that a participant is pregnant or may have been pregnant at the time of study exposure, including during at least 5 half-lives after product administration, the investigator must immediately notify the BMS Medical Monitor/designee of this event and complete and forward a Pregnancy Surveillance Form to BMS Designee within 24 hours of awareness of the event and in accordance with SAE reporting procedures described in Appendix 3

In most cases, the study treatment will be permanently discontinued in an appropriate manner (eg, dose tapering if necessary for participant safety). Please call the BMS Medical Monitor within 24 hours of awareness of the pregnancy.

Protocol-required procedures for study discontinuation and follow-up must be performed on the participant.

Any pregnancy that occurs in a female partner of a male study participant should be reported to Sponsor or designee. In order for Sponsor or designee to collect any pregnancy surveillance information from the female partner, the female partner must sign an informed consent form for disclosure of this information. Information on this pregnancy will be collected on the Pregnancy Surveillance Form.

# 9.2.6 Laboratory Test Result Abnormalities

The following laboratory test result abnormalities should be captured on the nonserious AE CRF page or SAE Report Form electronic, as appropriate. Paper forms are only intended as a back-up option when the electronic system is not functioning.

Any laboratory test result that is clinically significant or meets the definition of an SAE


37

- Any laboratory test result abnormality that required the participant to have study treatment discontinued or interrupted
- Any laboratory test result abnormality that required the participant to receive specific corrective therapy

It is expected that wherever possible, the clinical rather than laboratory term would be used by the reporting investigator (eg, anemia versus low hemoglobin value).

Some coagulation tests (eg, aPTT,) are affected by the investigational drug and therefore changes in such tests are not to be considered as AEs but as PD biomarkers.

# 9.2.7 Potential Drug Induced Liver Injury (DILI)

Wherever possible, timely confirmation of initial liver-related laboratory abnormalities should occur prior to the reporting of a potential DILI event. All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 9.2 and Appendix 3 for reporting details).

Potential drug induced liver injury is defined as:

Wherever possible, timely confirmation of initial liver-related laboratory abnormalities should occur prior to the reporting of a potential DILI event. All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Appendix 3 for reporting details).

Potential drug induced liver injury is defined as:

 AT (ALT or AST) elevation > 3 times ULN AND

 Total bilirubin > 2 times ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase),

AND

3) No other immediately apparent possible causes of AT elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic.

# 9.2.8 Other Safety Considerations

Any significant worsening noted during interim or final physical examinations, electrocardiogram, x-ray filming, any other potential safety assessment required or not required by protocol should also be recorded as a non-serious or serious AE, as appropriate, and reported accordingly.

### 9.3 Overdose

An overdose is defined as the accidental or intentional administration of any dose of a product that is considered both excessive and medically important. All occurrences of overdose must be reported as an SAE (see Section 9.2).

# 9.4 Safety

Planned timepoints for all safety assessments are listed in the Schedule of Activities.

# 9.4.1 Physical Examinations

Refer to Schedule of Activities.

# 9.4.2 Vital signs

Refer to Schedule of Activities.

# 9.4.3 Electrocardiograms

Refer to Schedule of Activities.

# 9.4.4 Clinical Safety Laboratory Assessments

Investigators must document their review of each laboratory safety report.

A local laboratory will perform the analyses and will provide reference ranges for these tests.

Results of clinical laboratory tests performed on Day -1 to -3 must be available prior to first dose of study drug.

| Hematology | |
|-----------------------------------------------|-----------------|
| Hemoglobin | |
| Hematocrit | |
| Total leukocyte count, including differential | |
| Platelet count | |
| Coagulation | |
| PT | |
| aPTT | |
| INR | |
| Serum Chemistry | |
| Aspartate aminotransferase (AST) | Total Protein |
| Alanine aminotransferase (ALT) | Albumin |
| Total bilirubin | Sodium |
| Direct bilirubin | Potassium |
| Alkaline phosphatase | Chloride |
| Lactate dehydrogenase (LDH) | Calcium |
| Creatinine | Phosphorus |
| Blood Urea Nitrogen (BUN) | Magnesium |
| Uric acid | Creatine kinase |
| Fasting glucose (if possible) | |

| Clinical Protocol | CV010010 |
|-------------------|----------|
| BMS-986177 | FXIa |

| Urine Dipstick |
|---|
| Blood (only if the participant is able to produce urine) |
| Serology |
| HIV-1 and -2 antibody (screening only) |
| Other Analyses |
| Test for drugs of abuse (urine or saliva or plasma) |
| Alcohol breathalyzer |
| Fecal occult blood (screening and after each treatment period if sample can be obtained) |
| Pregnancy test (urine or blood)- WOCBP only |

# 9.4.5 Suicidal Risk Monitoring

Not Applicable

# 9.4.6 Imaging Safety Assessment

Not Applicable

# 9.5 Pharmacokinetic

Pharmacokinetics of BMS-986177 will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include:

| Cmax | Maximum observed plasma concentration |
|---|---|
| Tmax | Time of maximum observed plasma concentration |
| AUC(0-T) | Area under the plasma concentration-time curve from time zero to time |
| | of last quantifiable concentration |
| AUC(INF) | Area under the plasma concentration-time curve from time zero |
| | extrapolated to infinite time |
| AUC(0-48) | Area under the plasma concentration-time curve from time zero to |
| | 48 hours |
| T-HALF | Terminal plasma half-life |
| fu | Fraction of unbound drug |
| Cmaxfu | Maximum observed plasma concentration of free drug |
| AUC(0-T)fu | Area under the plasma concentration-time curve from time zero to time |
| | of last quantifiable concentration of free drug |
| AUC(INF)fu | Area under the plasma concentration-time curve from time zero |
| | extrapolated to infinite time of free drug |
| AUC(3-7) | Area under the plasma concentration-time curve from 3 to 7 hours. (ie, |
| | during dialysis. Determined from blood samples entering and exiting the |
| | dialyzer) |
| %DR | Percent dose of BMS-986177 recovered in dialysate (%) |
| CLD | Dialysate clearance of drug from plasma |
| | Cumulative amount in dialysate over 3 to 7 hours postdose divided by |
| | plasma AUC(3-7) |

Individual participant pharmacokinetic parameter values will be derived by non-compartmental methods by a validated pharmacokinetic analysis program. Actual times will be used for the analyses.

Table 9.5-1: Pharmacokinetic Sampling Schedule for BMS-986177

| Day of Sample<br>Collection when<br>BMS-986177 is dosed | Event | Time<br>Relative to<br>BMS-986177<br>Dose)<br>Hour: Min | BMS-986177<br>Blood Sample<br>for PK | BMS-<br>986177<br>Protein<br>Binding<br>Sample | BMS-<br>986177<br>Dialysate<br>Sample |
|---|---|---|---|---|---|
| | predose | 00:00 | X <sup>a</sup> | | |
| | postdose | 1:00 | X | | |
| | hemodialysis<br>start <sup>c</sup> | 3:00 | x <sup>b</sup> | | |
| BMS-986177 dosing | | 3:30 | Xb | | |
| day (depending on randomization | | 4:00 | Xb | | X (3-7) <sup>e</sup> |
| sequence it may be<br>study day 1, 5, 8, or | | 5:00 | $X^{b}$ | X | |
| 12) | | 6:00 | $X^{b}$ | | |
| | hemodialysis<br>stop <sup>c</sup> | 7:00 | x <sup>b</sup> | | |
| | | 8:00 | X | | |
| | | 9:00 | X | | |
| 24 to 72 hours after<br>BMS-986177 dosing | | 24:00 - 72:00 <sup>d</sup> | х | | |

Note: Day 1, 5, 8, and 12 is the start of Period 1, 2, 3, and 4, respectively. Hemodialysis duration could range from 3 to 4 hours but should be consistent on the days when study drug is administered.

a Sample to be obtained prior to study drug administration.

Two blood samples are obtained at each of these time points (one sample is collected prior to entering the dialyzer and the second sample is collected after exiting the dialyzer) for Periods for BMS-986177 only

Sample to be collected from the blood prior to entering the dialyzer.

d Single sample between days 2-4, days 6-8, days 9-11, and days 13-15.

e Dialysate sample to be collected hourly between 3 to 7 hr during the hemodialysis session.

The plasma samples will be analyzed for BMS-986177 by a validated LC/MS/MS assay. In addition, plasma samples will be archived for potential metabolite analysis, if the need arises and to the extent possible.

Detailed instructions for the PK blood collection, labeling, processing, storage, and shipping will be provided to the site in the procedure manual.

After the scheduled PK analyses are completed, residual plasma may be used for metabolite profiling. If these analyses are conducted, they will be reported separately from the CSR.

# 9.6 Pharmacodynamics

BMS-986177

Blood will be drawn at the times indicated in Table 9.6-1 and Table 9.6-2, for the measurement of pharmacodynamic markers (PD): aPTT, and Factor XI clotting activity (FXIc) for BMS-986177, aPTT and Anti-Xa for heparin and Enoxaparin. Further details of blood collection and processing will be provided to the site in the procedure manual.

Table 9.6-1: Pharmacodynamic Sampling Schedule for dialysis session with BMS-986177 and Enoxaparin

| Event | Time<br>(Relative To BMS-BMS-<br>986177 or Enoxaparin<br>Dose )<br>Hour: Min | Blood Sample for aPTT,<br>FXIc<br>(BMS-986177 day only) <sup>a</sup> | Blood Sample for aPTT<br>and anti-Xa<br>(Enoxaparin day only) <sup>a</sup> |
|---|---|---|---|
| predose | 00:00 | X | X |
| | 01:00 | X | X |
| Hemodialysis start | 03:00 | x a | X a |
| | 04:00 | x a | X <sup>a</sup> |
| | 05:00 | x <sup>a</sup> | x a |
| | 06:00 | x <sup>a</sup> | x <sup>a</sup> |
| Hemodialysis stop | 07:00 | x a | x <sup>a</sup> |
| | 08:00 | X | X |
| | 09:00 | X | X |
| 24 to 72 hours after<br>BMS-986177 dosing | 24:00 - 72:00 <sup>b</sup> | Х | |

Note: Hemodialysis duration could range from 3 to 4 hours but should be consistent on the days when study drug is administered.

Revised Protocol No.: 03 Date: 06-Sep-2017 **FXIa** 

<sup>&</sup>lt;sup>a</sup> Blood sample is collected prior to entering the dialyzer.

b Single sample between days 2-4, days 6-8, days 9-11, and days 13-15.

| Table 9.6-2: Pharmacodynamic Sampling Schedule for dialysis session with UFH | <b>Table 9.6-2:</b> | Pharmacodynamic Sa | ampling Schedule for | dialysis session with UFH |
|---|---|---|---|---|
|---|---|---|---|---|

| Event | Time<br>(Relative To UFH Dose )<br>Hour: Min | Blood Sample for aPTT and anti-Xa<br>(UFH days only) |
|---|---|---|
| Predose/ Hemodialysis start | 00:00 | X <sup>a</sup> |
| | 01:00 | X <sup>a</sup> |
| | 02:00 | X <sup>a</sup> |
| | 03:00 | X <sup>a</sup> |
| Hemodialysis stop | 04:00 | X <sup>a</sup> |
| | 05:00 | Х |
| | 06:00 | X |

Note: Hemodialysis duration could range from 3 to 4 hours but should be consistent on the days when study drug is administered.

# 9.7 Pharmacogenomics

BMS-986177

# 9.7.1 Genotyping and ADME Sampling

A 6-mL whole blood sample will be drawn at baseline for dosed participants as indicated in Section 2 Schedule of Activities) for potential analysis of DNA variants in ADME-related genes (see Appendix 5) which contains the lists of ADME-related genes from http://pharmaadme.org), and/or hemostasis and thrombosis related genes. Further details of blood collection and processing will be provided to the site in the procedure manual.



Revised Protocol No.: 03 Date: 06-Sep-2017 **FXIa** 

<sup>&</sup>lt;sup>a</sup> Blood sample is collected prior to entering the dialyzer.

MS- 86177 Factor XIa In

Clinical Protocol CV010010 BMS-986177 FXIa



### 9.8.1 Additional Research Collection

Additional research collections and retention are mandatory for all subjects, except where prohibited by local laws or regulations.

This protocol will include residual sample storage for additional research (AR).

This collection for additional research is intended to expand the translational R&D capability at Bristol-Myers Squibb, and will support as yet undefined research aims that will advance our understanding of disease and options for treatment. It may also be used to support health authority requests for analysis, and advancement of pharmacodiagnostic development to better target drugs to the right patients. This may also include genetic/genomic exploration aimed at exploring disease pathways, progression and response to treatment etc.

All requests for access to samples or data for additional research will be vetted through a diverse committee of the study sponsor's senior leaders in Research and Development to ensure the research supports appropriate and well-defined scientific research activities.

Residual plasma from PD and biomarker collections (see Table 9.6-1, Table 9.6-2, Table 9.8-1, and Table 9.8-2) will also be retained for additional research purposes.

Samples will be securely stored by the BMS Biorepository in NJ or at a BMS approved third party storage management facility.

Samples will be stored in a coded fashion, and no researcher will have access to the key. The key is securely held by the Investigator at the clinical site, so there is no direct ability for a researcher to connect a sample to a specific individual

Additional research samples will be retained for 15 years or the maximum allowed by applicable law. No additional sampling is required for residual collections.

Further details of sample collection and processing will be provided to the site in the procedure manual.

Table 9.8.1-1: Residual Sample Retention for Additional Research Schedule

| Sample Type | Timepoints for which residual samples will be retained |
|---|---|
| D-dimer, F1.2 and exploratory sample | All time points as in Table 9.8-1 and Table 9.8-2 |
| aPTT, FXIc, anti-Xa | All time points as in Table 9.6-1 and Table 9.6-2 |

### 9.8.2 Other Assessments

Not Applicable

#### 9.9 Health Economics OR Medical Resource Utilization and Health **Economics**

Health Economics/Medical Resource Utilization and Health Economics parameters will not be evaluated in this study.

#### 10. STATISTICAL CONSIDERATIONS

#### 10.1 Sample Size Determination

Although the number of patients is not based on statistical power considerations, administration of BMS-986177 to 32 subjects with ESRD would provide over 80% probability of observing at least one occurrence of any adverse event that would occur with incidence of 5% in the population from which the sample is drawn

#### 10.2 **Populations for Analyses**

For purposes of analysis, the following populations are defined:

| Population | Description |
|---|---|
| Enrolled | All subjects who sign informed consent |
| Randomized | All subjects who are randomized to the study including the subjects who replace the discontinuing randomized subjects |
| Evaluable | All randomized subjects who take at least 1 dose of study treatment. |
| Safety | All randomized subjects who take at least 1 dose of study treatment. |
| Pharmacokinetic | All participants who receive BMS-986177 from whom PK parameter data were obtained before and after HD. |
| Pharmacodynamic | Is a subset of the Safety Population and includes all subjects who received at least 1 dose of study medication and had any available PD or biomarker data. |

#### 10.3 Statistical Analyses

The statistical analysis plan will be developed and finalized before database lock and will describe the selection of participants to be included in the analyses, and procedures for accounting for missing, unused, and spurious data. Below is a summary of planned statistical analyses of the primary and secondary endpoints.


**FXIa** 

| o- 801// | Factor Ata III |
|-------------------|----------------|
| Clinical Protocol | CV010010 |
| BMS-986177 | FXIa |

# 10.3.1 Efficacy Analyses

| Endpoint | Statistical Analysis Methods |
|----------|------------------------------|
| Primary | NA |

# 10.3.2 Safety Analyses

Safety analyses will be performed on all safety assessments.

| Endpoint | Statistical Analysis Methods |
|---|---|
| Primary | Descriptive summaries will be presented for continuous variables using number of subjects (N), mean, standard deviation (SD), median, minimum and maximum. Descriptive summaries for categorical variables will utilize counts and percentages. |
| | All recorded AEs will be listed and tabulated by system organ class and preferred term, and treatment. Changes from baseline in vital signs, ECG, and clinical laboratory test results will be listed and summarized by treatment and time point. Any significant physical examination findings and any marked abnormal clinical laboratory test results will be listed. Electrocardiogram readings will be summarized by time point, and investigator-identified abnormalities, if present, will be listed. |

# 10.3.3 Pharmacokinetic Analyses

| Endpoint | Statistical Analysis Methods |
|---|---|
| See section | Descriptive summaries will be presented for continuous variables using |
| 9.5 for all PK | number of subjects (N), mean, standard deviation (SD), median, minimum |
| parameters | and maximum. Geometric mean and coefficient of variation (%CV) will also |
| | be presented for sample plasma concentration-time data and PK parameters. |



| Final Clinical Study Report | CV010010 |
|-----------------------------|---------------|
| MS- 86177 | Factor XIa In |
| Clinical Protocol | CV010010 |
| BMS-986177 | FXIa |

Results of DNA variants and other exploratory measures may not be reported in the CSR.

# 10.3.5 Interim Analyses

Not Applicable

| Final Clinical Study Report | CV010010 |
|-----------------------------|---------------|
| MS- 86177 | Factor XIa In |
| Clinical Protocol | CV010010 |
| BMS-986177 | FXIa |

# 12 APPENDICES

Clinical Protocol BMS-986177

CV010010 FXIa

# APPENDIX 1 ABBREVIATIONS AND TRADEMARKS

| Term | Definition |
|---|---|
| ADME | Absorption, distribution, metabolism, excretion |
| AE | adverse event |
| ACLS | advanced cardiac life support |
| ALT | alanine aminotransferase |
| ANC | absolute neutrophil count |
| aPTT | activated partial thromboplastin time |
| ARIC | Atherosclerosis Risk in Communities |
| AST | aspartate aminotransferase |
| AT | aminotransaminases |
| AUC | area under the concentration-time curve |
| AUC(INF) | area under the concentration-time curve from time zero extrapolated to infinite time |
| AUC(0-T) | area under the concentration-time curve from time zero to the time of the last quantifiable concentration |
| AUC(TAU) | area under the concentration-time curve in one dosing interval |
| β-HCG | beta-human chorionic gonadotrophin |
| BID, bid | bis in die, twice daily |
| BLQ | below limit of quantification |
| BMI | body mass index |
| BMS | Bristol-Myers Squibb |
| BP | blood pressure |
| BUN | blood urea nitrogen |
| С | Celsius |
| Ca <sup>++</sup> | calcium |
| CBC | complete blood count |
| CFR | Code of Federal Regulations |
| CI | confidence interval |
| C1- | chloride |
| CLcr | creatinine clearance |
| CLD | Dialysate clearance of drug from plasma/serum |

MS- 86177

Clinical Protocol BMS-986177 CV010010 FXIa

| Term | Definition |
|---|---|
| cm | centimeter |
| Cmax, CMAX | maximum observed concentration |
| Cmin, CMIN | minimum observed concentration |
| CNS | Central nervous system |
| CONSORT | Consolidated Standards of Reporting Trials |
| CRC | Clinical Research Center |
| CRF | Case Report Form, paper or electronic |
| CV | coefficient of variation |
| СҮР | cytochrome p-450 |
| D/C | discontinue |
| dL | deciliter |
| DMC | Data monitoring committee |
| DRt, DR | Total amount recovered in dialysate |
| %DRt, %DR | Total percent of administered dose recovered in dialysate |
| DSM IV | Diagnostic and Statistical Manual of Mental Disorders (4 <sup>th</sup> Edition) |
| DVT | deep vein thrombosis |
| EC20, EC50,<br>EC80 | Effective concentration at 20%, 50%, 80% |
| ECG | electrocardiogram |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| eg, e.g. | exempli gratia (for example) |
| ESR | Expedited Safety Report |
| ESRD | end-stage renal disease |
| F | bioavailability |
| FIH | First in human |
| FDA | Food and Drug Administration |
| FSH | follicle stimulating hormone |
| fu | fraction of unbound drug |
| FXI | Factor XI |
| FXIa | Factor XIa |

Factor XIa In

MS- 86177 Clinical Protocol

BMS-986177

CV010010 FXIa

| Term | Definition |
|---|---|
| FXIc | Factor XI clotting activity |
| g | gram |
| GC | gas chromatography |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transferase |
| h | hour |
| HBsAg | hepatitis B surface antigen |
| HBV | hepatitis B virus |
| HCV | hepatitis C virus |
| HCO <sub>3</sub> - | bicarbonate |
| HD | hemodialysis |
| HIT | heparin-induced thrombocytopenia |
| HIV | Human Immunodeficiency Virus |
| HR | heart rate |
| HRT | hormone replacement therapy |
| IB | investigator brochure |
| ICD | International Classification of Diseases |
| ICH | International Conference on Harmonisation |
| ie, i.e. | id est (that is) |
| IEC | Independent Ethics Committee |
| IMP | investigational medicinal products |
| IND | Investigational New Drug Exemption |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| IU | International Unit |
| IUD | intrauterine devices |
| IV, I.V. | intravenous |
| K | slope of the terminal phase of the log concentration-time curve |
| K <sub>3</sub> EDTA | potassium ethylenediaminetetraacetic acid |
| K <sup>+</sup> | potassium |

Factor XIa In

MS- 86177

Clinical Protocol BMS-986177 CV010010 FXIa

| Term | Definition |
|---|---|
| Ki | inhibition constant |
| kg | kilogram |
| Kt/V | Number used to quantify hemodialysis and peritoneal dialysis treatment adequacy. Assessment includes: pre-dialysis blood BUN, post-dialysis blood BUN, ultrafiltration volume, post-dialysis body weight, duration of dialysis session. |
| L | liter |
| LAM | lactation amenorrhea method |
| LC | liquid chromatography |
| LDH | lactate dehydrogenase |
| LFTs | liver function tests |
| LMWH | low molecular weight heparin |
| MAD | multiple ascending dose |
| mg | milligram |
| Mg <sup>++</sup> | magnesium |
| min | minute |
| mL | milliliter |
| mmHg | millimeters of mercury |
| MR | medical research |
| MS | mass spectrometry |
| μg | microgram |
| N | number of subjects or observations |
| Na <sup>+</sup> | sodium |
| N/A, NA | not applicable |
| ng | nanogram |
| NIMP | non-investigational medicinal products |
| NOAEL | no-observed-adverse-effect-level |
| NSAID | nonsteroidal anti-inflammatory drug |
| P2Y12 | Gi class of a group of G protein-coupled (GPCR) purinergic receptors and is a chemoreceptor for adenosine diphosphate (ADP) |
| PD | pharmacodynamics |

MS- 86177

Clinical Protocol BMS-986177 CV010010 FXIa

| Term | Definition |
|---|---|
| PID | patient identification number |
| PK | pharmacokinetics |
| PO | per os (by mouth route of administration) |
| PT | prothrombin time |
| PTT | partial thromboplastin time |
| QC | quality control |
| QD, qd | quaque die, once daily |
| RATIO | Risk of Arterial Thrombosis In relation to Oral contraceptives |
| RBC | red blood cell |
| SAD | single ascending dose |
| SAE | serious adverse event |
| SC | subcutaneous |
| SD | standard deviation |
| SDD | spray dry dispersion |
| SOA | schedule of activities |
| SOC | standard of care |
| SOP | Standard Operating Procedures |
| t | temperature |
| Т | time |
| TAO | Trial Access Online, the BMS implementation of an EDC capability |
| T-HALF | Half life |
| TID, tid | ter in die, three times a day |
| Tmax, TMAX | time of maximum observed concentration |
| UFH | unfractionated heparin |
| ULN | upper limit of normal |
| WBC | white blood cell |
| WHO | World Health Organization |
| WOCBP | women of childbearing potential |
| WNOCBP | women <u>not</u> of childbearing potential |
| х д | times gravity |

# BMS-986177

#### STUDY GOVERANCE CONSIDERATIONS **APPENDIX 2**

The term 'Participant' is used in the protocol to refer to a person who has consented to participate in the clinical research study. The term 'Subject' used in the eCRF is intended to refer to a person (Participant) who has consented to participate in the clinical research study.

# REGULATORY AND ETHICAL CONSIDERATIONS **GOOD CLINICAL PRACTICE**

This study will be conducted in accordance with:

- Good Clinical Practice (GCP),
- as defined by the International Council on Harmonisation (ICH)
- in accordance with the ethical principles underlying European Union Directive 2001/20/EC
- United States Code of Federal Regulations, Title 21, Part 50 (21CFR50)
- applicable local requirements.

The study will be conducted in compliance with the protocol. The protocol and any amendments and the participant informed consent will receive approval/favorable opinion by Institutional Review Board/Independent Ethics Committee (IRB/IEC), and regulatory authorities according to applicable local regulations prior to initiation of the study.

All potential serious breaches must be reported to Sponsor or designee immediately. A serious breach is a breach of the conditions and principles of GCP in connection with the study or the protocol, which is likely to affect, to a significant degree, the safety or physical or mental integrity of the subjects of the study or the scientific value of the study.

Personnel involved in conducting this study will be qualified by education, training, and experience to perform their respective tasks.

This study will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (e.g., loss of medical licensure, debarment).

### INSTITUTIONAL REVIEW BOARD/INDEPENDENT ETHICS COMMITTEE

Before study initiation, the investigator must have written and dated approval/favorable opinion from the IRB/IEC for the protocol, consent form, participant recruitment materials (e.g., advertisements), and any other written information to be provided to subjects. The investigator or BMS should also provide the IRB/IEC with a copy of the Investigator Brochure or product labeling information to be provided to subjects and any updates.

The investigator, Sponsor or designee should provide the IRB/IEC with reports, updates and other information (e.g., expedited safety reports, amendments, and administrative letters) according to regulatory requirements or institution procedures.

## COMPLIANCE WITH THE PROTOCOL AND PROTOCOL REVISIONS

The investigator should not implement any deviation or change to the protocol without prior review and documented approval/favorable opinion of an amendment from the IRB/IEC (and if applicable, also by local health authority) except where necessary to eliminate an immediate hazard(s) to study subjects.

If a deviation or change to a protocol is implemented to eliminate an immediate hazard(s) prior to obtaining relevant approval/favorable opinion(s) the deviation or change will be submitted, as soon as possible to:

- IRB/IEC for
- Regulatory Authority(ies), if applicable by local regulations (per national requirements)

Documentation of approval/favorable opinion signed by the chairperson or designee of the IRB(s)/IEC(s) and if applicable, also by local health authority must be sent to BMS.

If an amendment substantially alters the study design or increases the potential risk to the participant: (1) the consent form must be revised and submitted to the IRB(s)/IEC(s) for review and approval/favorable opinion; (2) the revised form must be used to obtain consent from subjects currently enrolled in the study if they are affected by the amendment; and (3) the new form must be used to obtain consent from new subjects prior to enrollment.

If the revision is done via an administrative letter, investigators must inform their IRB(s)/IEC(s).

# FINANCIAL DISCLOSURE

Investigators and sub-Investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate health authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

### INFORMED CONSENT PROCESS

Investigators must ensure that subjects are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which they volunteer to participate.

In situations where consent cannot be given to subjects, their legally acceptable representatives (as per country guidelines) are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which the participant volunteers to participate.

Sponsor or designee will provide the investigator with an appropriate (i.e., Global or Local) sample informed consent form which will include all elements required by ICH, GCP and applicable regulatory requirements. The sample informed consent form will adhere to the ethical principles that have their origin in the Declaration of Helsinki.

Investigators must:


60

- Provide a copy of the consent form and written information about the study in the language in which the participant is most proficient prior to clinical study participation. The language must be non-technical and easily understood.
- Allow time necessary for participant or participant's legally acceptable representative to inquire about the details of the study.
- Obtain an informed consent signed and personally dated by the participant or the participant's legally acceptable representative and by the person who conducted the informed consent discussion.
- Obtain the IRB/IEC's written approval/favorable opinion of the written informed consent form and any other information to be provided to the subjects, prior to the beginning of the study, and after any revisions are completed for new information.

If informed consent is initially given by a participant's legally acceptable representative or legal guardian, and the participant subsequently becomes capable of making and communicating his or her informed consent during the study, consent must additionally be obtained from the participant.

Revise the informed consent whenever important new information becomes available that is relevant to the participant's consent. The investigator, or a person designated by the investigator, should fully inform the participant or the participant's legally acceptable representative or legal guardian, of all pertinent aspects of the study and of any new information relevant to the participant's willingness to continue participation in the study. This communication should be documented.

The confidentiality of records that could identify subjects must be protected, respecting the privacy and confidentiality rules applicable to regulatory requirements, the subjects' signed ICF and, in the US, the subjects' signed HIPAA Authorization.

The consent form must also include a statement that BMS and regulatory authorities have direct access to participant records.

The rights, safety, and well-being of the study subjects are the most important considerations and should prevail over interests of science and society.

### SOURCE DOCUMENTS

The Investigator is responsible for ensuring that the source data are accurate, legible, contemporaneous, original and attributable, whether the data are hand-written on paper or entered electronically. If source data are created (first entered), modified, maintained, archived, retrieved, or transmitted electronically via computerized systems (and/or any other kind of electronic devices) as part of regulated clinical trial activities, such systems must be compliant with all applicable laws and regulations governing use of electronic records and/or electronic signatures. Such systems may include, but are not limited to, electronic medical/health records

(EMRs/EHRs), adverse event tracking/reporting, protocol required assessments, and/or drug accountability records).

When paper records from such systems are used in place of electronic format to perform regulated activities, such paper records should be certified copies. A certified copy consists of a copy of original information that has been verified, as indicated by a dated signature, as an exact copy having all of the same attributes and information as the original.

# STUDY TREATMENT RECORDS

Records for study treatments (whether supplied by BMS, its vendors, or the site) must substantiate study treatment integrity and traceability from receipt, preparation, administration, and through destruction or return. Records must be made available for review at the request of BMS/designee or a Health Authority.

| If | Then |
|---|---|
| Supplied by BMS (or its vendors): | Records or logs must comply with applicable |
| | regulations and guidelines and should |
| | include: |
| | amount received and placed in storage |
| | area |
| | amount currently in storage area |
| | label identification number or batch<br>number |
| | <ul> <li>amount dispensed to and returned by each<br/>participant, including unique participant<br/>identifiers</li> </ul> |
| | amount transferred to another area/site for dispensing or storage |
| | • nonstudy disposition (e.g., lost, wasted) |
| | amount destroyed at study site, if applicable |
| | amount returned to BMS |
| | retain samples for<br>bioavailability/bioequivalence, if<br>applicable |
| | dates and initials of person responsible for<br>Investigational Product<br>dispensing/accountability, as per the<br>Delegation of Authority Form. |
| Sourced by site, and not supplied by BMS or | The investigator or designee accepts |
| its vendors (examples include IP sourced | responsibility for documenting traceability |
| from the sites stock or commercial supply, or | and study drug integrity in accordance with |
| | requirements applicable under law and the |

Clinical Protocol BMS-986177 CV010010 FXIa

| If | Then |
|---|---|
| a specialty pharmacy) | SOPs/standards of the sourcing pharmacy. |
| | These records should include: |
| | label identification number or batch<br>number |
| | amount dispensed to and returned by each participant, including unique participant identifiers |
| | dates and initials of person responsible for<br>Investigational Product<br>dispensing/accountability, as per the<br>Delegation of Authority Form. |

BMS or designee will provide forms to facilitate inventory control if the investigational site does not have an established system that meets these requirements.

### CASE REPORT FORMS

An investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the investigation on each individual treated or entered as a control in the investigation. Data that are derived from source documents and reported on the CRF must be consistent with the source documents or the discrepancies must be explained. Additional clinical information may be collected and analyzed in an effort to enhance understanding of product safety. CRFs may be requested for AEs and/or laboratory abnormalities that are reported or identified during the course of the study.

For sites using the Sponsor or designee electronic data capture tool, electronic CRFs will be prepared for all data collection fields except for fields specific to SAEs and pregnancy, which will be reported on the electronic SAE form and Pregnancy Surveillance form, respectively. If electronic SAE form is not available, a paper SAE form can be used. Spaces may be left blank only in those circumstances permitted by study-specific CRF completion guidelines provided by Sponsor or designee.

The confidentiality of records that could identify subjects must be protected, respecting the privacy and confidentiality rules in accordance with the applicable regulatory requirement(s).

The investigator will maintain a signature sheet to document signatures and initials of all persons authorized to make entries and/or corrections on CRFs.

The completed CRF, SAE/pregnancy CRFs, must be promptly reviewed, signed, and dated by the investigator or qualified physician who is a subinvestigator and who is delegated this task on the Delegation of Authority Form. Subinvestigators in Japan may not be delegated the CRF approval For electronic CRFs, review and approval/signature is completed electronically through the BMS electronic data capture tool. The investigator must retain a copy of the CRFs including records of the changes and corrections.

Each individual electronically signing electronic CRFs must meet Sponsor or designee training requirements and must only access the BMS electronic data capture tool using the unique user account provided by Sponsor or designee. User accounts are not to be shared or reassigned to other individuals

# MONITORING

Sponsor or designee representatives will review data centrally to identify potential issues to determine a schedule of on-site visits for targeted review of study records.

Representatives of BMS must be allowed to visit all study site locations periodically to assess the data quality and study integrity. On site they will review study records and directly compare them with source documents, discuss the conduct of the study with the investigator, and verify that the facilities remain acceptable Certain CRF pages and/or electronic files may serve as the source documents:

In addition, the study may be evaluated by Sponsor or designee internal auditors and government inspectors who must be allowed access to CRFs, source documents, other study files, and study facilities. BMS audit reports will be kept confidential.

The investigator must notify BMS promptly of any inspections scheduled by regulatory authorities, and promptly forward copies of inspection reports to Sponsor or designee.

# **RECORDS RETENTION**

The investigator (or head of the study site in Japan) must retain all study records and source documents for the maximum period required by applicable regulations and guidelines, or institution procedures, or for the period specified by BMS or designee, whichever is longer. The investigator (or head of the study site in Japan) must contact BMS prior to destroying any records associated with the study.

BMS or designee will notify the investigator (or head of the study site in Japan) when the study records are no longer needed.

If the investigator withdraws from the study (e.g., relocation, retirement), the records shall be transferred to a mutually agreed upon designee (e.g., another investigator, study site, IRB). Notice of such transfer will be given in writing to BMS or designee.

# RETURN OF STUDY TREATMENT

For this study, study treatments (those supplied by BMS, a vendor or sourced by the investigator) such as partially used study treatment containers, vials and syringes may be destroyed on site.

| If | Then |
|---|---|
| Study treatments supplied by BMS (including | Any unused study treatments supplied by |
| its vendors | BMS can only be destroyed after being |
| | inspected and reconciled by the responsible |
| | Study Monitor unless study treatments |
| | containers must be immediately destroyed as |

| Clinical Protocol | CV010010 |
|-------------------|----------|
| BMS-986177 | FXIa |

| | required for safety, or to meet local regulations (e.g., cytotoxics or biologics). |
|---|---|
| | If study treatments will be returned, the return will be arranged by the responsible Study Monitor. |
| by BMS (or its vendors) (examples include | It is the investigator's or designee's responsibility to dispose of all containers according to the institutional guidelines and procedures. |

It is the investigator's or designee's responsibility to arrange for disposal, provided that procedures for proper disposal have been established according to applicable federal, state, local, and institutional guidelines and procedures, and provided that appropriate records of disposal are kept. The following minimal standards must be met:

- On-site disposal practices must not expose humans to risks from the drug.
- On-site disposal practices and procedures are in agreement with applicable laws and regulations, including any special requirements for controlled or hazardous substances.
- Written procedures for on-site disposal are available and followed. The procedures must be filed with the site's SOPs and a copy provided to BMS upon request.
- Records are maintained that allow for traceability of each container, including the date disposed of, quantity disposed, and identification of the person disposing the containers.
   The method of disposal, i.e., incinerator, licensed sanitary landfill, or licensed waste disposal vendor must be documented.
- Accountability and disposal records are complete, up-to-date, and available for the Monitor to review throughout the clinical trial period.

It is the investigator's or designee's responsibility to arrange for disposal of all empty containers.

If conditions for destruction cannot be met the responsible Study Monitor will make arrangements for return of study treatments provided by BMS (or its vendors). Destruction of non-study treatments sourced by the site, not supplied by BMS, is solely the responsibility of the investigator or designee.

It is however, the investigator's or designee's responsibility to arrange for disposal of all empty study treatment containers, provided that procedures for proper disposal have been established according to applicable federal, state, local, and institutional guidelines and procedures, and provided that appropriate records of disposal are kept. The return of full or partially used study treatments supplied by BMS or its vendors will be arranged by the responsible Study Monitor.

# **CLINICAL STUDY REPORT AND PUBLICATIONS**

A Signatory Investigator must be selected to sign the clinical study report.

For this protocol, the Signatory Investigator will be selected as appropriate based on the following criteria:

- · External Principal Investigator designated at protocol development
- Participant recruitment (e.g., among the top quartile of enrollers)
- Involvement in trial design
- Other criteria (as determined by the study team)

The data collected during this study are confidential and proprietary to Sponsor or designee. Any publications or abstracts arising from this study must adhere to the publication requirements set forth in the clinical trial agreement (CTA) governing [Study site or Investigator] participation in the study. These requirements include, but are not limited to, submitting proposed publications to Sponsor or designee at the earliest practicable time prior to submission or presentation and otherwise within the time period set forth in the CTA.

APPENDIX 3 ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS: DEFINITIONS AND PROCEDURES FOR RECORDING, EVALUATING, FOLLOW UP AND REPORTING

### **ADVERSE EVENTS**

### **Adverse Event Definition:**

An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.

## SERIOUS ADVERSE EVENTS

# Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose:

# Results in death

Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)

Requires inpatient hospitalization or causes prolongation of existing hospitalization (see NOTE below)

## NOTE:

The following hospitalizations are not considered SAEs in BMS clinical studies:

- a visit to the emergency room or other hospital department < 24 hours, that does not result in admission (unless considered an important medical or lifethreatening event)
- o elective surgery, planned prior to signing consent
- o admissions as per protocol for a planned medical/surgical procedure
- routine health assessment requiring admission for baseline/trending of health status (e.g., routine colonoscopy)
- o medical/surgical admission other than to remedy ill health and planned prior to entry into the study. Appropriate documentation is required in these cases
- admission encountered for another life circumstance that carries no bearing on health status and requires no medical/surgical intervention (e.g., lack of housing, economic inadequacy, caregiver respite, family circumstances, administrative reason)
- admission for administration of anticancer therapy in the absence of any other SAEs (applies to oncology protocols)

Results in persistent or significant disability/incapacity

Is a congenital anomaly/birth defect

is an important medical event (defined as a medical event(s) that may not be immediately life-threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the participant or may require intervention [e.g., medical, surgical] to prevent one of the other serious outcomes listed in the definition above.) Examples of such events include, but are not limited to, intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization.) Potential drug induced liver injury (DILI) is also considered an important medical event. (See Section 8.1.1 for the definition of potential DILI.)

Suspected transmission of an infectious agent (e.g., pathogenic or nonpathogenic) via the study treatment is an SAE.

Although pregnancy, overdose, cancer, and potential drug induced liver injury (DILI) are not always serious by regulatory definition, these events must be handled as SAEs. (See Section 9.2.5 for reporting pregnancies).

Any component of a study endpoint that is considered related to study therapy should be reported as SAE (e.g., death is an endpoint, if death occurred due to anaphylaxis, anaphylaxis must be reported).

## **EVALUATING AES AND SAES**

# Assessment of Causality

The causal relationship to study drug is determined by a physician and should be used to assess all adverse events (AE). The causal relationship can be one of the following:

Related: There is a reasonable causal relationship between study drug administration and the AE.

Not related: There is not a reasonable causal relationship between study drug administration and the AE.

The term "reasonable causal relationship" means there is evidence to suggest a causal relationship.

# Follow-up of AEs and SAEs

If only limited information is initially available, follow-up reports are required. (Note: Follow-up SAE reports must include the same investigator term(s) initially reported.)

If an ongoing SAE changes in its intensity or relationship to study drug or if new information becomes available, the SAE report must be updated and submitted within 24 hours to BMS (or designee) using the same procedure used for transmitting the initial SAE report.

All SAEs must be followed to resolution or stabilization.

# REPORTING OF SAES TO SPONSOR OR DESIGNEE

- SAEs, whether related or not related to study drug, and pregnancies must be reported to BMS (or designee) within 24 hours of awareness of the event.
- SAEs must be recorded on the SAE Report Form; pregnancies on a Pregnancy Surveillance Form (electronic or paper forms).
- The preferred method for SAE data reporting collection is through the eCRF.
- The paper SAE/pregnancy surveillance forms are only intended as a back-up option when the eCRF system is not functioning.
  - In this case, the paper forms are to be transmitted via email or confirmed facsimile (fax) transmission to:

SAE Email Address: Refer to Contact Information list.

# SAE Facsimile Number: Refer to Contact Information list.

For studies capturing SAEs through electronic data capture (EDC), electronic submission is the required method for reporting. In the event the electronic system is unavailable for transmission, paper forms must be used and submitted immediately. When paper forms are used, the original paper forms are to remain on site.

SAE Telephone Contact (required for SAE and pregnancy reporting): Refer to Contact Information list

BMS-986177 **FXIa** 

#### **APPENDIX 4** WOMEN OF CHILDBEARING POTENTIAL DEFINITIONS AND METHODS OF CONTRACEPTION

### DEFINITIONS

# Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

# Women in the following categories are not considered WOCBP

- Premenarchal
- Premenopausal female with 1 of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.

- Postmenopausal female
  - A postmenopausal state is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.

Note: Females treated with hormone replacement therapy, (HRT) are likely to have artificially suppressed FSH levels and may require a washout period in order to obtain a physiologic FSH level. The duration of the washout period is a function of the type of HRT used. The duration of the washout period below are suggested guidelines and the investigators should use their judgement in checking serum FSH levels.

- 1 week minimum for vaginal hormonal products (rings, creams, gels)
- 4 week minimum for transdermal products
- 8 week minimum for oral products

Other parenteral products may require washout periods as long as 6 months. If the serum FSH level is > 40 mIU/ml at any time during the washout period, the woman can be considered postmenopausal.

# CONTRACEPTION GUIDANCE FOR FEMALE PARTICIPANTS OF CHILD BEARING **POTENTIAL**

Any one of the approved methods of contraception (highly effective and/or less than highly effective) listed below is required during study duration plus 5 half-lives of study treatment


71

BMS-986177 FXIa

BMS-986177 (2 days) plus 30 days (duration of ovulatory cycle) for a total of 32 days post-treatment completion or after treatment has been discontinued.

Local laws and regulations may require use of alternative and/or additional contraception methods.

# Table 1-1: Methods of Contraception

### Highly Effective Contraceptive Methods That Are User Dependent

Failure rate of <1% per year when used consistently and correctly.<sup>a</sup>

- Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation<sup>b</sup>
  - oral
  - intravaginal
  - transdermal
- Progestogen-only hormonal contraception associated with inhibition of ovulation<sup>b</sup>
  - oral
  - injectable

## Highly Effective Methods That Are User Independent

- Implantable progestogen-only hormonal contraception associated with inhibition of ovulation <sup>b</sup>
- Intrauterine device (IUD)<sup>c</sup>
- Intrauterine hormone-releasing system (IUS)<sup>c</sup>
- Bilateral tubal occlusion

### Vasectomized partner

A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

### Sexual abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

- It is not necessary to use any other method of contraception when complete abstinence is elected.
- WOCBP participants who choose complete abstinence must continue to have pregnancy tests, as specified in Section 2.
- Acceptable alternate methods of highly effective contraception must be discussed in the event that the WOCBP participants chooses to forego complete abstinence

### Less Than Highly Effective Contraceptive Methods That Are User Dependent

Failure rate of >1% per year when used consistently and correctly.

- Male or female condom with or without spermicide. Male and female condoms cannot be used simultaneously
- · Diaphragm with spermicide
- · Cervical cap with spermicide
- Vaginal Sponge with spermicide


644
## Table 1-1: Methods of Contraception

 Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mechanism of action

#### **Unacceptable Methods of Contraception**

- Periodic abstinence (calendar, symptothermal, post-ovulation methods)
- Withdrawal(coitus interruptus).
- · Spermicide only
- Lactation amenorrhea method (LAM)

#### NOTES:

- <sup>a</sup> Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies.
- b Hormonal contraception may be susceptible to interaction with the study treatment, which may reduce the efficacy of the contraceptive method. Hormonal contraception is permissible only when there is sufficient evidence that the IMP and other study medications will not alter hormonal exposures such that contraception would be ineffective or result in increased exposures that could be potentially hazardous. In this case, hormonal methods of contraception can be utilized.
- Intrauterine devices and intrauterine hormone releasing systems are acceptable methods of contraception in the absence of definitive drug interaction studies when hormone exposures from intrauterine devices do not alter contraception effectiveness

# CONTRACEPTION GUIDANCE FOR MALE PARTICIPANTS WITH PARTNER(S) OF CHILD BEARING POTENTIAL.

Male participants with female partners of childbearing potential are eligible to participate if they agree to the following during the treatment and until the end of relevant systemic exposure.

- Inform any and all partner(s) of their participation in a clinical drug study and the need to comply with contraception instructions as directed by the investigator.
- Male participants are required to use a condom for study duration and until the end of relevant systemic exposure defined as 2 days after the end of treatment in the male participant with amendment/revised protocol 02 (See Section 6.1 Inclusion Criteria).
- Female partners of males participating in the study to consider use of effective methods of contraception (see Table 1-1) until the end of relevant systemic exposure, defined as 2 days after the end of treatment in the male participant.
- Male participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile vaginal intercourse or use a male condom during each episode of penile penetration during the treatment and until 2 days after the end of treatment.
- Refrain from donating sperm for the duration of the study treatment and for 2 days after the end of treatment with amendment/revised protocol 02 (See Section 6.1 Inclusion Criteria).

| Final Clinical Study Report | CV010010 |
|-----------------------------|---------------|
| MS- 86177 | Factor XIa In |
| Clinical Protocol | CV010010 |
| BMS-986177 | FXIa |

#### **COLLECTION OF PREGNANCY INFORMATION**

Guidance for collection of Pregnancy Information and outcome of pregnancy on the Pregnancy Surveillance Form is provided in Section 9.2.5 and the Appendix for Adverse Events and Serious Adverse Events Definitions and procedures for Evaluating, Follow-up and Reporting.

Clinical Protocol BMS-986177 CV010010 FXIa

## APPENDIX 5 CORE ADME GENE LIST (FROM HTTP://PHARMAADME.ORG)

| Gene<br>Symbol | Full Gene Name | Class |
|---|---|---|
| ABCB1 | ATP-binding cassette, sub-family B (MDR/TAP), member 1 | Transporter |
| ABCC2 | ATP-binding cassette, sub-family C (CFTR/MRP), member $2$ | Transporter |
| ABCG2 | ATP-binding cassette, sub-family G (WHITE), member 2 | Transporter |
| CYP1A1 | cytochrome P450, family 1, subfamily A, polypeptide 1 | Phase I |
| CYP1A2 | cytochrome P450, family 1, subfamily A, polypeptide 2 | Phase I |
| CYP2A6 | cytochrome P450, family 2, subfamily A, polypeptide 6 | Phase I |
| CYP2B6 | cytochrome P450, family 2, subfamily B, polypeptide 6 | Phase I |
| CYP2C19 | cytochrome P450, family 2, subfamily C, polypeptide 19 | Phase I |
| CYP2C8 | cytochrome P450, family 2, subfamily C, polypeptide 8 | Phase I |
| CYP2C9 | cytochrome P450, family 2, subfamily C, polypeptide 9 | Phase I |
| CYP2D6 | cytochrome P450, family 2, subfamily D, polypeptide 6 | Phase I |
| CYP2E1 | cytochrome P450, family 2, subfamily E, polypeptide 1 | Phase I |
| CYP3A4 | cytochrome P450, family 3, subfamily A, polypeptide 4 | Phase I |
| CYP3A5 | cytochrome P450, family 3, subfamily A, polypeptide 5 | Phase I |
| DPYD | dihydropyrimidine dehydrogenase | Phase I |
| GSTM1 | glutathione S-transferase M1 | Phase II |
| GSTP1 | glutathione S-transferase pi | Phase II |
| GSTT1 | glutathione S-transferase theta 1 | Phase II |
| NAT1 | N-acetyltransferase 1 (arylamine N-acetyltransferase) | Phase II |
| NAT2 | N-acetyltransferase 2 (arylamine N-acetyltransferase) | Phase II |
| SLC15A2 | solute carrier family 15 (H+/peptide transporter), member 2 | Transporter |
| SLC22A1 | solute carrier family 22 (organic cation transporter), member 1 | Transporter |
| SLC22A2 | solute carrier family 22 (organic cation transporter), member 2 | Transporter |
| SLC22A6 | solute carrier family 22 (organic anion transporter), member 6 | Transporter |
| SLCO1B1 | solute carrier organic anion transporter family, member 1B1 | Transporter |
| SLCO1B3 | solute carrier organic anion transporter family, member 1B3 | Transporter |
| SULT1A1 | sulfotransferase family, cytosolic, 1A, phenol-preferring, member1 | Phase II |
| TPMT | thiopurine S-methyltransferase, | Phase II |

Clinical Protocol CV010010 BMS-986177 FXIa

| Gene<br>Symbol | Full Gene Name | Class |
|---|---|---|
| UGT1A1 | UDP glucuronosyltransferase 1 family, polypeptide A1 | Phase II |
| UGT2B15 | UDP glucuronosyltransferase 2 family, polypeptide B15 | Phase II |
| UGT2B17 | UDP glucuronosyltransferase 2 family, polypeptide B17 | Phase II |
| UGT2B7 | UDP glucuronosyltransferase 2 family, polypeptide B7 | Phase II |

## **EXTENDED ADME GENE LIST:**

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| ABCB8 | ATP-binding cassette, sub-family B (MDR/TAP), member 8 | Transporter |
| ABCC12 | ATP-binding cassette, sub-family C (CFTR/MRP), member 12 | Transporter |
| ABCC3 | ATP-binding cassette, sub-family C (CFTR/MRP), member $3$ | Transporter |
| ABCC4 | ATP-binding cassette, sub-family C (CFTR/MRP), member 4 | Transporter |
| AHR | aryl hydrocarbon receptor | Modifier |
| ALDH4A1 | aldehyde dehydrogenase 4 family, member A1 | Phase I |
| ALDH5A1 | aldehyde dehydrogenase 5 family, member A1 | Phase I |
| ALDH6A1 | aldehyde dehydrogenase 6 family, member A1 | Phase I |
| CES1 | carboxylesterase 1 (monocyte/macrophage serine esterase 1) | Phase I |
| CES2 | carboxylesterase 2 (intestine, liver) | Phase I |
| CYP7A1 | cytochrome P450, family 7, subfamily A, polypeptide 1 | Phase I |
| EPHX1 | epoxide hydrolase 1, microsomal (xenobiotic) | Phase I |
| FMO3 | flavin containing monooxygenase 3 | Phase I |
| GSTA1 | glutathione S-transferase A1 | Phase II |
| GSTA2 | glutathione S-transferase A2 | Phase II |
| GSTA3 | glutathione S-transferase A3 | Phase II |
| GSTA4 | glutathione S-transferase A4 | Phase II |
| GSTA5 | glutathione S-transferase A5 | Phase II |
| GSTM2 | glutathione S-transferase M2 (muscle),glutathione S-transferase M4 | Phase II |
| GSTM3 | glutathione S-transferase M3 (brain) | Phase II |
| GSTM4 | glutathione S-transferase M4 | Phase II |
| GSTO1 | glutathione S-transferase omega 1,glutathione S-transferase omega 2 | Phase II |
| GSTO2 | glutathione S-transferase omega 2 | Phase II |
| GSTT2 | glutathione S-transferase theta 2 | Phase II |
| SLC10A1 | solute carrier family 10 (sodium/bile acid cotransporter family),<br>member 1 | Transporter |

Clinical Protocol CV010010 BMS-986177 FXIa

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| SLC15A1 | solute carrier family 15 (oligopeptide transporter), member 1 | Transporter |
| SLC22A11 | solute carrier family 22 (organic anion/cation transporter), member 11 | Transporter |
| SLC22A8 | solute carrier family 22 (organic anion transporter), member 8 | Transporter |
| SLC7A5 | solute carrier family 7 (cationic amino acid transporter, y+ system), member 5 | Transporter |
| SLCO1A2 | solute carrier organic anion transporter family, member 1A2 | Transporter |
| SLCO2B1 | solute carrier organic anion transporter family, member 2B1 | Transporter |
| SULT1A2 | sulfotransferase family, cytosolic, 1A, phenol-preferring, member 2 | Phase II |
| SULT1A3 | sulfotransferase family, cytosolic, 1A, phenol-preferring, member 3 | Phase II |
| SULT1B1 | sulfotransferase family, cytosolic, 1B, member 1 | Phase II |
| UGT1A3 | UDP glucuronosyltransferase 1 family, polypeptide A3 | Phase II |
| UGT1A6 | UDP glucuronosyltransferase 1 family, polypeptide A6 | Phase II |
| UGT1A7 | UDP glucuronosyltransferase 1 family, polypeptide A7 | Phase II |
| UGT1A8 | UDP glucuronosyltransferase 1 family, polypeptide A8 | Phase II |
| UGT1A9 | UDP glucuronosyltransferase 1 family, polypeptide A9 | Phase II |
| UGT2A1 | UDP glucuronosyltransferase 2 family, polypeptide A1 | Phase II |
| UGT2B11 | UDP glucuronosyltransferase 2 family, polypeptide B11 | Phase II |
| UGT2B28 | UDP glucuronosyltransferase 2 family, polypeptide B28 | Phase II |
| UGT2B4 | UDP glucuronosyltransferase 2 family, polypeptide B4 | Phase II |
| ABCA1 | ATP-binding cassette, sub-family A (ABC1), member 1 | Transporter |
| ABCA4 | ATP-binding cassette, sub-family A (ABC1), member 4 | Transporter |
| ABCB11 | ATP-binding cassette, sub-family B (MDR/TAP), member 11 | Transporter |
| ABCB4 | ATP-binding cassette, sub-family B (MDR/TAP), member 4 | Transporter |
| ABCB5 | ATP-binding cassette, sub-family B (MDR/TAP), member 5 | Transporter |
| ABCB6 | ATP-binding cassette, sub-family B (MDR/TAP), member 6 | Transporter |

Clinical Protocol BMS-986177 CV010010 FXIa

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| ABCB7 | ATP-binding cassette, sub-family B (MDR/TAP), member 7 | Transporter |
| ABCC1 | ATP-binding cassette, sub-family C (CFTR/MRP), member 1 | Transporter |
| ABCC10 | ATP-binding cassette, sub-family C (CFTR/MRP), member 10 | Transporter |
| ABCC11 | ATP-binding cassette, sub-family C (CFTR/MRP), member 11 | Transporter |
| ABCC5 | ATP-binding cassette, sub-family C (CFTR/MRP), member 5 | Transporter |
| ABCC6 | ATP-binding cassette, sub-family C (CFTR/MRP), member 6 | Transporter |
| ABCC8 | ATP-binding cassette, sub-family C (CFTR/MRP), member 8 | Transporter |
| ABCC9 | ATP-binding cassette, sub-family C (CFTR/MRP), member 9 | Transporter |
| ABCG1 | ATP-binding cassette, sub-family G (WHITE), member 1 | Transporter |
| ADH1A | alcohol dehydrogenase 1A (class I), alpha polypeptide | Phase I |
| ADH1B | alcohol dehydrogenase IB (class I), beta polypeptide | Phase I |
| ADH1C | alcohol dehydrogenase 1C (class I), gamma polypeptide | Phase I |
| ADH4 | alcohol dehydrogenase 4 (class II), pi polypeptide | Phase I |
| ADH5 | alcohol dehydrogenase 5 (class III), chi polypeptide,<br>methionyl<br>aminopeptidase 1 | Phase I |
| ADH6 | alcohol dehydrogenase 6 (class V) | Phase I |
| ADH7 | alcohol dehydrogenase 7 (class IV), mu or sigma polypeptide | Phase I |
| ALDH1A1 | aldehyde dehydrogenase 1 family, member A1 | Phase I |
| ALDH1A2 | aldehyde dehydrogenase 1 family, member A2 | Phase I |
| ALDH1A3 | aldehyde dehydrogenase 1 family, member A3 | Phase I |
| ALDH1B1 | aldehyde dehydrogenase 1 family, member B1 | Phase I |
| ALDH2 | aldehyde dehydrogenase 2 family (mitochondrial) | Phase I |
| ALDH3A1 | aldehyde dehydrogenase 3 family, memberA1 | Phase I |
| ALDH3A2 | aldehyde dehydrogenase 3 family, member A2 | Phase I |
| ALDH3B1 | aldehyde dehydrogenase 3 family, member B1 | Phase I |
| ALDH3B2 | aldehyde dehydrogenase 3 family, member B2 | Phase I |

Factor XIa In

MS- 86177
Clinical Protocol

BMS-986177

CV010010 FXIa

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| ALDH7A1 | aldehyde dehydrogenase 7 family, member A1 | Phase I |
| ALDH8A1 | aldehyde dehydrogenase 8 family, member A1 | Phase I |
| ALDH9A1 | aldehyde dehydrogenase 9 family, member A1 | Phase I |
| AOX1 | aldehyde oxidase 1 | Phase I |
| ARNT | aryl hydrocarbon receptor nuclear translocator | Modifier |
| CBR1 | carbonyl reductase 1 | Phase I |
| CBR3 | carbonyl reductase 3 | Phase I |
| CDA | cytidine deaminase | Modifier |
| CYB5R3 | cytochrome b5 reductase 3 | Phase I |
| CYP11A1 | cytochrome P450, family 11, subfamily A, polypeptide 1 | Phase I |
| CYP11B1 | cytochrome P450, family 11, subfamily B, polypeptide 1 | Phase I |
| CYP11B2 | cytochrome P450, family 11, subfamily B, polypeptide 2 | Phase I |
| CYP17A1 | cytochrome P450, family 17, subfamily A, polypeptide 1 | Phase I |
| CYP1B1 | cytochrome P450, family 1, subfamily B, polypeptide 1 | Phase I |
| CYP20A1 | cytochrome P450, family 20, subfamily A, polypeptide 1 | Phase I |
| CYP20A1 | cytochrome P450, family 20, subfamily A, polypeptide 1 | Phase I |
| CYP21A2 | cytochrome P450, family 21, subfamily A, polypeptide 2 | Phase I |
| CYP24A1 | cytochrome P450, family 24, subfamily A, polypeptide 1 | Phase I |
| CYP26A1 | cytochrome P450, family 26, subfamily A, polypeptide 1 | Phase I |
| CYP27A1 | cytochrome P450, family 27, subfamily A, polypeptide 1 | Phase I |
| CYP2A13 | cytochrome P450, family 2, subfamily A, polypeptide 13 | Phase I |
| CYP2A7 | cytochrome P450, family 2, subfamily A, polypeptide 7 | Phase I |
| CYP2C18 | cytochrome P450, family 2, subfamily C, polypeptide 18 | Phase I |
| CYP2F1 | cytochrome P450, family 2, subfamily F, polypeptide 1 | Phase I |
| CYP2J2 | cytochrome P450, family 2, subfamily J, polypeptide 2 | Phase I |
| CYP39A1 | cytochrome P450, family 39, subfamily A, polypeptide 1 | Phase I |
| CYP3A43 | cytochrome P450, family 3, subfamily A, polypeptide 43 | Phase I |
| CYP3A7 | cytochrome P450, family 3, subfamily A, polypeptide 7 | Phase I |
| CYP4B1 | cytochrome P450, family 4, subfamily B, polypeptide 1 | Phase I |
| CYP4F11 | cytochrome P450, family 4, subfamily F, polypeptide 11 | Phase I |
| CYP51A1 | cytochrome P450, family 51, subfamily A, polypeptide 1 | Phase I |
| EPHX2 | epoxide hydrolase 2, cytoplasmic | Phase I |
| FMO1 | flavin containing monooxygenase 1 | Phase I |
| FMO2 | flavin containing monooxygenase 2 | Phase I |

Clinical Protocol CV010010 BMS-986177 FXIa

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| FMO4 | flavin containing monooxygenase 4 | Phase I |
| FMO5 | flavin containing monooxygenase 5 | Phase I |
| GPX2 | glutathione peroxidase 2 (gastrointestinal) | Phase I |
| GPX3 | glutathione peroxidase 3 (plasma) | Phase I |
| GPX7 | glutathione peroxidase 7 | Phase I |
| GSR | glutathione reductase | Phase I |
| GSTK1 | glutathione S-transferase kappa 1 | Phase II |
| GSTM5 | glutathione S-transferase M5 | Phase II |
| GSTZ1 | glutathione transferase zeta 1 (maleylacetoacetate isomerase) | Phase II |
| NNMT | nicotinamide N-methyltransferase | Phase II |
| NR1I2 | nuclear receptor subfamily 1, group I, member 2 | Modifier |
| NR1I3 | nuclear receptor subfamily 1, group I, member 3 | Modifier |
| PNMT | phenylethanolamine N-methyltransferase | Phase II |
| PON1 | paraoxonase 1 | Phase I |
| PON2 | paraoxonase 2 | Phase I |
| PON3 | paraoxonase 3 | Phase I |
| POR | P450 (cytochrome) oxidoreductase | Modifier |
| PPARD | peroxisome proliferative activated receptor, delta | Modifier |
| PPARG | peroxisome proliferative activated receptor, gamma | Modifier |
| RXRA | retinoid X receptor, alpha | Modifier |
| SLC10A2 | solute carrier family 10 (sodium/bile acid cotransporter family), member 2 | Transporter |
| SLC13A1 | solute carrier family 13 (sodium/sulfate symporters), member 1 | Transporter |
| SLC13A2 | solute carrier family 13 (sodium-dependent dicarboxylate transporter), member 2 | Transporter |
| SLC13A3 | solute carrier family 13 (sodium-dependent dicarboxylate transporter), member 3 | Transporter |
| SLC16A1 | solute carrier family 16 (monocarboxylic acid Transporter), member 1 | Transporter |
| SLC19A1 | solute carrier family 19 (folate transporter), member 1 | Transporter |

Clinical Protocol CV010010 BMS-986177 FXIa

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| SLC22A10 | solute carrier family 22 (organic anion/cation transporter), member 10 | Transporter |
| SLC22A12 | solute carrier family 22 (organic anion/cation transporter), member 12 | Transporter |
| SLC22A13 | solute carrier family 22 (organic cation transporter), member 13 | Transporter |
| SLC22A14 | solute carrier family 22 (organic cation transporter), member 14 | Transporter |
| SLC22A15 | solute carrier family 22 (organic cation transporter), member 15 | Transporter |
| SLC22A16 | solute carrier family 22 (organic cation transporter), member 16 | Transporter |
| SLC22A17 | solute carrier family 22 (organic cation transporter), member 17 | Transporter |
| SLC22A18 | solute carrier family 22 (organic cation transporter), member 18 | Transporter |
| SLC22A18AS | solute carrier family 22 (organic cation transporter),<br>member 18<br>antisense | Transporter |
| SLC22A3 | solute carrier family 22 (extraneuronal monoamine transporter), member 3 | Transporter |
| SLC22A4 | solute carrier family 22 (organic cation transporter), member 4 | Transporter |
| SLC22A5 | solute carrier family 22 (organic cation transporter), member 5 | Transporter |
| SLC22A7 | solute carrier family 22 (organic anion transporter), member 7 | Transporter |
| SLC22A9 | solute carrier family 22 (organic anion/cation transporter), member 9 | Transporter |
| SLC27A1 | solute carrier family 27 (fatty acid transporter), member 1 | Transporter |
| SLC28A1 | solute carrier family 28 (sodium-coupled nucleoside transporter), member 1 | Transporter |
| SLC28A2 | solute carrier family 28 (sodium-coupled nucleoside transporter), member 2 | Transporter |

Clinical Protocol CV010010 BMS-986177 FXIa

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| SLC28A3 | solute carrier family 28 (sodium-coupled nucleoside transporter), member 3 | Transporter |
| SLC29A1 | solute carrier family 29 (nucleoside Transporter), member 1 | Transporter |
| SLC29A2 | solute carrier family 29 (nucleoside Transporter), member 2 | Transporter |
| SLC2A4 | solute carrier family 2 (facilitated glucose transporter), member 4 | Transporter |
| SLC2A5 | solute carrier family 2 (facilitated glucose/fructose transporter), member 5 | Transporter |
| SLC5A6 | solute carrier family 5 (sodium-dependent vitamin transporter) | Transporter |
| SLC6A6 | solute carrier family 6 (neurotransmitter transporter, taurine), member 6 | Transporter |
| SLC7A8 | solute carrier family 7 (cationic amino acid transporter, y+ system), member 8 | Transporter |
| SLCO1C1 | solute carrier organic anion transporter family, member 1C1 | Transporter |
| SLCO2A1 | solute carrier organic anion transporter family, member 2A1 | Transporter |
| SLCO3A1 | solute carrier organic anion transporter family, member 3A1 | Transporter |
| SLCO4A1 | solute carrier organic anion transporter family, member 4A1 | Transporter |
| SLCO4C1 | solute carrier organic anion transporter family, member 4C1 | Transporter |
| SLCO5A1 | solute carrier organic anion transporter family, member 5A1 | Transporter |
| SLCO6A1 | solute carrier organic anion transporter family, member 6A1 | Transporter |
| SULT1C1 | sulfotransferase family, cytosolic, 1C, member 1 | Phase II |
| SULT1C2 | sulfotransferase family, cytosolic, 1C, member 2 | Phase II |
| SULT1E1 | sulfotransferase family 1E, estrogen-preferring, member 1 | Phase II |

Clinical Protocol BMS-986177 CV010010 FXIa

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| SULT2A1 | sulfotransferase family, cytosolic, 2A, DHEA preferring, member 1 | Phase II |
| SULT2B1 | sulfotransferase family, cytosolic, 2B, member 1 | Phase II |
| TAP1 | transporter 1, ATP-binding cassette, sub-family B (MDR/TAP) | Transporter |
| UGT1A10 | UDP glucuronosyltransferase 1 family, polypeptide A10 | Phase II |
| UGT1A4 | UDP glucuronosyltransferase 1 family, polypeptide A4 | Phase II |
| UGT1A5 | UDP glucuronosyltransferase 1 family, polypeptide A5 | Phase II |
| UGT2B10 | UDP glucuronosyltransferase 2 family, polypeptide B10 | Phase II |
| ABCC13 | ATP-binding cassette, sub-family C (CFTR/MRP), member 13 | Transporter |
| ARSA | arylsulfatase A | Modifier |
| CAT | catalase | Modifier |
| CHST8 | carbohydrate (N-acetylgalactosamine 4-0) sulfotransferase 8 | Phase II |
| CYP19A1 | cytochrome P450, family 19, subfamily A, polypeptide 1 | Phase I |
| CYP26C1 | cytochrome P450, family 26, subfamily C, polypeptide 1 | Phase I |
| CYP27B1 | cytochrome P450, family 27, subfamily B, polypeptide 1 | Phase I |
| CYP2R1 | cytochrome P450, family 2, subfamily R, polypeptide 1 | Phase I |
| CYP2S1 | cytochrome P450, family 2, subfamily S, polypeptide 1 | Phase I |
| CYP46A1 | cytochrome P450, family 46, subfamily A, polypeptide 1 | Phase I |
| CYP4A11 | cytochrome P450, family 4, subfamily A, polypeptide 11 | Phase I |
| CYP4F12 | cytochrome P450, family 4, subfamily F, polypeptide 12 | Phase I |
| CYP4F2 | cytochrome P450, family 4, subfamily F, polypeptide 2 | Phase I |
| CYP4F3 | cytochrome P450, family 4, subfamily F, polypeptide 3 | Phase I |
| CYP4F8 | cytochrome P450, family 4, subfamily F, polypeptide 8 | Phase I |
| CYP4Z1 | cytochrome P450, family 4, subfamily Z, polypeptide 1 | Phase I |
| CYP7B1 | cytochrome P450, family 7, subfamily B, polypeptide 1 | Phase I |
| CYP8B1 | cytochrome P450, family 8, subfamily B, polypeptide 1 | Phase I |
| DHRS13 | dehydrogenase/reductase (SDR family) member 13 | Phase I |
| DHRS2 | dehydrogenase/reductase (SDR family) member 2 | Phase I |
| GPX1 | glutathione peroxidase 1 | Phase I |
| GPX4 | glutathione peroxidase 4 (phospholipid hydroperoxidase) | Phase I |
| GPX5 | glutathione peroxidase 5 (epididymal androgen-related protein) | Phase I |

Clinical Protocol BMS-986177 CV010010 FXIa

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| GPX6 | glutathione peroxidase 6 (olfactory) | Phase I |
| GSS | glutathione synthetase | Phase I |
| GSTCD | glutathione S-transferase, C-terminal domain containing | Phase II |
| HNF4A | hepatocyte nuclear factor 4, alpha | Modifier |
| HNMT | histamine N-methyltransferase | Phase II |
| HSD11B1 | hydroxysteroid (17-beta) dehydrogenase 11 | Phase I |
| HSD17B11 | hydroxysteroid (17-beta) dehydrogenase 11 | Phase I |
| HSD17B14 | hydroxysteroid (17-beta) dehydrogenase 14 | Phase I |
| LOC731356 | similar to dehydrogenase/reductase (SDR family) member 4 like 2 | Phase I |
| MGST1 | microsomal glutathione S-transferase 1 | Phase II |
| MGST2 | microsomal glutathione S-transferase 2 | Phase II |
| MGST3 | microsomal glutathione S-transferase 3 | Phase II |
| MPO | myeloperoxidase | Modifier |
| NOS1 | nitric oxide synthase 1 (neuronal) | Phase I |
| NOS2A | nitric oxide synthase 2A (inducible, hepatocytes) | Phase I |
| NOS3 | nitric oxide synthase 3 (endothelial cell) | Phase I |
| PPARA | peroxisome proliferator-activated receptor alpha | Modifier |
| SERPINA7 | serpin peptidase inhibitor, clade A (alpha-1 antiproteinase, antitrypsin), member 7 | Modifier |
| SLC7A7 | solute carrier family 7 (cationic amino acid transporter, y+system), member 7 | Transporter |
| SOD1 | superoxide dismutase 1, soluble (amyotrophic lateral sclerosis 1 [adult]) | Modifier |
| SOD2 | superoxide dismutase 2, mitochondrial | Modifier |
| SOD3 | superoxide dismutase 3, extracellular precursor | Modifier |
| SULF1 | sulfatase 1 | Phase I |
| SULT4A1 | sulfotransferase family 4A, member 1 | Phase II |
| TAP2 | transporter 2, ATP-binding cassette, sub-family B (MDR/TAP) | Transporter |
| UGT8 | UDP glycosyltransferase 8 (UDP-galactose ceramide galactosyltransferase) | Phase II |

Clinical Protocol BMS-986177 CV010010 FXIa

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| XDH | xanthine dehydrogenase | Phase I |
| ADHFE1 | alcohol dehydrogenase, iron containing, 1 | Phase I |
| CHST1 | carbohydrate (keratan sulfate Gal-6) sulfotransferase 1 | Phase II |
| CHST10 | carbohydrate sulfotransferase 10 | Phase II |
| CHST11 | carbohydrate (chondroitin 4) sulfotransferase 11 | Phase II |
| CHST12 | carbohydrate (chondroitin 4) sulfotransferase 12 | Phase II |
| CHST13 | carbohydrate (chondroitin 4) sulfotransferase 13 | Phase II |
| CHST2 | carbohydrate (N-acetylglucosamine-6-O) sulfotransferase 2 | Phase II |
| CHST3 | carbohydrate (chondroitin 6) sulfotransferase 3 | Phase II |
| CHST4 | carbohydrate (N-acetylglucosamine 6-O) sulfotransferase 4 | Phase II |
| CHST5 | carbohydrate (N-acetylglucosamine 6-O) sulfotransferase 5 | Phase II |
| CHST6 | carbohydrate (N-acetylglucosamine 6-O) sulfotransferase 6 | Phase II |
| CHST7 | carbohydrate (N-acetylglucosamine 6-O) sulfotransferase 7 | Phase II |
| CHST9 | carbohydrate (N-acetylgalactosamine 4-0) sulfotransferase 9 | Phase II |
| CYP2D7P1 | cytochrome P450, family 2, subfamily D, polypeptide 7 pseudogene 1 | Phase I |
| DDO | D-aspartate oxidase | Phase I |
| DHRS1 | dehydrogenase/reductase (SDR family) member 1 | Phase I |
| DHRS12 | dehydrogenase/reductase (SDR family) member 12 | Phase I |
| DHRS3 | dehydrogenase/reductase (SDR family) member 3 | Phase I |
| DHRS4 | dehydrogenase/reductase (SDR family) member 4 | Phase I |
| DHRS4L1 | dehydrogenase/reductase (SDR family) member 4 like 1 | Phase I |
| DHRS4L2 | dehydrogenase/reductase (SDR family) member 4 like 2 | Phase I |
| DHRS7 | dehydrogenase/reductase (SDR family) member 7 | Phase I |
| DHRS7B | dehydrogenase/reductase (SDR family) member 7B | Phase I |
| DHRS7C | dehydrogenase/reductase (SDR family) member 7C | Phase I |
| DHRS9 | dehydrogenase/reductase (SDR family) member 9 | Phase I |
| DHRSX | dehydrogenase/reductase (SDR family) X-linked | Phase I |
| DPEP1 | dipeptidase 1 (renal) | Phase I |

CV010010

- 86177 Factor XIa In

Clinical Protocol

BMS-986177 CV010010

FXIa

| Gene Symbol | Full Gene Name | Class |
|---|---|---|
| FMO6P | flavin containing monooxygenase 6 | Phase I |
| HAGH | hydroxyacylglutathione hydrolase | Phase I |
| IAPP | islet amyloid polypeptide | Modifier |
| KCNJ11 | potassium inwardly-rectifying channel, subfamily J, member 11 | Modifier |
| LOC728667 | similar to dehydrogenase/reductase (SDR family) member 2 isoform 1 | Phase I |
| LOC731931 | similar to dehydrogenase/reductase (SDR family) member 2 isoform 1 | Phase I |
| MAT1A | methionine adenosyltransferase I, alpha | Modifier |
| METAP1 | methionyl aminopeptidase 1 | Phase I |
| PDE3A | phosphodiesterase 3A, cGMP-inhibited | Phase I |
| PDE3B | phosphodiesterase 3B, cGMP-inhibited | Phase I |
| PLGLB1 | plasminogen-like B1 | Phase I |
| ATP7A | ATPase, Cu++ transporting, alpha polypeptide (Menkes syndrome) | Modifier |
| ATP7B | ATPase, Cu++ transporting, beta polypeptide | Modifier |
| CFTR | cystic fibrosis transmembrane conductance regulator | Modifier |

# APPENDIX 6 DIAGNOSTIC CRITERIA FOR DRUG AND ALCOHOL ABUSE

The following is taken from DSM-IV:

BMS-986177

#### Diagnostic Criteria for Psychoactive Substance Dependence

A maladaptive pattern of substance use, leading to clinically significant impairment or distress as manifested by three (or more) of the following, occurring at any time in the same 12-month period:

- 1. Tolerance, as defined by either of the following:
  - a) A need for markedly increased amounts of the substance to achieve intoxication or desired effect.
  - b) Markedly diminished effect with continued use of the same amount of the substance.
- 2. Withdrawal, as manifested by either of the following:
  - a) The characteristic withdrawal syndrome for the substance,
  - b) The same (or closely related) substance is taken to relieve or avoid withdrawal symptoms.
- 3. The substance is often taken in larger amounts or over a longer period than was intended.
- 4. There is a persistent desire or unsuccessful efforts to cut down or control substance use.
- 5. A great deal of time is spent in activities necessary to obtain the substance (eg, visiting multiple doctors or driving long distances), use the substance (eg, chain-smoking) or recover from its effects.
- 6. Important social, occupational or recreational activities are given up or reduced because of substance use.
- 7. The substance use is continued despite knowledge of having a persistent or recurring physical or psychological problem that is likely to have been caused or exacerbated by the substance (eg, current cocaine use despite recognition of cocaine-induce depression, or continued drinking despite recognition that an ulcer was made worse by alcohol consumption.)

Criteria for Severity of Psychoactive Substance Dependence:

Mild: Few, if any, symptoms in excess of those required to make the diagnosis, and the symptoms result in no more than mild impairment in occupational functioning or in usual social activities or relationships with others.

Moderate: Symptoms or functional impairment between "mild" and "severe".

Severe: Many symptoms in excess of those required to make the diagnosis, and the symptoms markedly interfere with occupational functioning or with usual social activities or relationships with others.

In Partial Remission: During the past six months, some use of the substance and some symptoms of dependence.


88

**FXIa** 

| Final Clinical Study Report | CV010010 |
|-----------------------------|---------------|
| MS- 86177 | Factor XIa In |
| Clinical Protocol | CV010010 |

BMS-986177 FXIa

In Full Remission: During the past six months, either no use of the substance, or use of the

# Diagnostic Criteria for Psychoactive Substance Abuse

substance and no symptoms of dependence.

- A. A maladaptive pattern of psychoactive substance use, leading to clinically significant impairment or distress as manifested by one (or more) of the following, occurring at any time in the same 12-month period:
  - Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (e.g., repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school, neglect of children or household).
  - 2. Recurrent substance use in situations in which it is physically hazardous (eg, driving an automobile or operating a machine when impaired by substance use).
  - 3. Recurrent substance-related legal problems (eg, arrests for substance-related disorderly conduct).
  - 4. Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (eg, arguments with spouse about consequences of intoxication, physical fights).
- B. The symptoms have never met the criteria for substance dependence for this class of substance.

Clinical Protocol CV010010 BMS-986177 FXIa



| SUMMARY OF KEY CHANGES OF REVISED PROTOCOL 02 | |
|---|---|
| Section Number<br>& Title | Description of Change |
| Title Page | Updated study director/medical monitor. |
| 2 Schedule of<br>Activities (SOA) | Duplicate row for pregnancy test was deleted and the Day 8 pregnancy test was moved to Day 13 to 15/Study Discharge column and clarified for WOCBP only. Clarified vital signs, stool occult blood, whole blood for genotyping/ADME, and SAEs. |
| 2 SOA and 9.4.4<br>Clinical Safety<br>Laboratory<br>Assessments | Clarified urine dipstick for blood only if the participant is able to produce urine. Clarified that the pregnancy test is for WOCBP only. |
| 2 Schedule of<br>Activities (SOA)<br>5.1 Overall<br>Design | Updated the screening window from 21 days to 28 days. |
| 5.2 Number of<br>Participants | Clarified the target sample size of 32 participants is to achieve 24 participants who complete the 4 study treatments. |

CV010010 FXIa

| SUMMARY OF KEY CHANGES OF REVISED PROTOCOL 02 | |
|---|---|
| Section Number<br>& Title | Description of Change |
| 6.2 Exclusion<br>Criteria | Clarify prior aspirin use to at least 1 week before dosing in exclusion criteria 2a. Updated duration contraceptive methods to be used for men in exclusion criteria 3e. |
| 7.7.1 Prohibited<br>and/or Restricted<br>Treatments | Clarify concomitant use of NSAIDS or aspirin to within 1 week prior to study drug administration. Also allow the use of topical antifungals. |
| 9.5<br>Pharmacokinetics | Extraction ratio was deleted |
| 9.7.1 Genotyping<br>and ADME<br>Sampling | Clarify that whole blood sample to be drawn at baseline for dosed participants. |
| Appendix 4 WOCBP Definitions and Methods of Contraception | Requirements for WOCBP participants to use one highly effective and/or one less effective method of contraceptive has been added. Duration of contraceptive methods for males has been updated to align with updating exclusion criteria 3e. |
| Title Page | Updated study director/medical monitor. |
| 2 Schedule of<br>Activities (SOA) | Duplicate row for pregnancy test was deleted and the Day 8 pregnancy test was moved to Day 13 to 15/Study Discharge column and clarified for WOCBP only. Clarified vital signs, stool occult blood, whole blood for genotyping/ADME, and SAEs. |

MS- 86177

Clinical Protocol BMS-986177 CV010010 FXIa

| SUMMARY OF KEY CHANGES OF REVISED PROTOCOL 02 | | |
|---|---|---|
| Section Number<br>& Title | Description of Change | Brief Rationale |
| 2 SOA and 9.4.4<br>Clinical Safety<br>Laboratory<br>Assessments | Clarified urine dipstick for blood only if the participant is able to produce urine. Clarified that the pregnancy test is for WOCBP only. | Clarification added based on feedback<br>from a site that many of the end stage<br>renal disease patients (ESRD) are<br>unable to produce urine. |
| 2 Schedule of<br>Activities (SOA)<br>5.1 Overall<br>Design | Updated the screening window from 21 days to 28 days. | Being a hemodialysis patient study, flexible in the screening period is needed to schedule the study with the participant's hemodialysis schedule. |
| 5.2 Number of<br>Participants | Clarified the target sample size of 32 participants is to achieve 24 participants who complete the 4 study treatments. | It was not intended to achieve 24 evaluable participants as previously written which would be those who received 1 dose of study drug. |
| 6.2 Exclusion<br>Criteria | Clarify prior aspirin use to at least 1 week before dosing in exclusion criteria 2a. Updated duration contraceptive methods to be used for men in exclusion criteria 3e. | Updated based on review of screen failures and the change will not likely impact the study assessment or patient safety. Definitive embryo-fetal development (EFD) studies have been completed and findings from these studies indicate that BMS-986177 is non-terogenic and non-genotoxic. |
| 7.7.1 Prohibited<br>and/or Restricted<br>Treatments | Clarify concomitant use of NSAIDS or aspirin to within 1 week prior to study drug administration. Also allow the use of topical antifungals. | Updated based on review of screen failures. These changes will not likely impact the study assessment or patient safety. |
| 9.5<br>Pharmacokinetics | Extraction ratio was deleted | It was a duplication to %DR (Percent dose of BMS-986177 recovered in dialysate %). |
| 9.7.1 Genotyping<br>and ADME<br>Sampling | Clarify that whole blood sample to be drawn at baseline for dosed participants. | To make this consistent with Section 2<br>Schedule of Activities (SOA). |
| Appendix 4 WOCBP Definitions and Methods of Contraception | Requirements for WOCBP participants to use one highly effective and/or one less effective method of contraceptive has been added. Duration of contraceptive | Appendix has been updated to reflect the latest protocol model template. Definitive embryo-fetal development (EFD) studies have been completed and findings from these studies indicate that BMS-986177 is non-terogenic and non- |

| SUMMARY OF KEY CHANGES OF REVISED PROTOCOL 02 | | |
|---|---|---|
| Section Number<br>& Title | Description of Change | Brief Rationale |
| | methods for males has been<br>updated to align with updating<br>exclusion criteria 3e. | genotoxic. |


BMS-986177

FXIa

Clinical Protocol

BMS-986177

MS- 86177

CV010010 FXIa



| SUMMARY OF KEY CHANGES FOR REVISED PROTOCOL 01 | |
|---|---|
| Section Number<br>& Title | Description of Change |
| Section 3.3:<br>Benefit/Risk<br>Assessment | Safety data was updated from FIH SAD/MAD study (CV010001). Also, the safety data from the HD PK study (CV010012) was added. |
| Section 5.1:<br>Overall Design | BMS dose 1 and BMS dose 2<br>were updated to be BMS-<br>986177 100 mg and BMS-<br>986177 300 mg, respectively. |
| | Other minor changes made in this section. |
| Section 5.5:<br>Justification for<br>Dose | Updated targeted exposures<br>based on hemodialysis PK<br>study to support the BMS<br>dose 1 (100 mg) and BMS<br>dose 2 (300 mg) |
| Section 6.2:<br>Exclusion Criteria<br>and Section 6.3:<br>Lifestyle<br>Restrictions | Exclusion criteria 1a, 1d, 1i, 1n, 3b, and 3e were clarified. Exclusion criterion 2b was added. Restrictions were updated. |
| Section 7:<br>Treatment | BMS-986177 100 mg and 300 mg (to replace BMS dose 1 and dose 2) were added to Table 7.1-1 and Table 7.1-1. |
| Section 7.2:<br>Method of<br>Treatment | Reference to IRT was removed. |

MS- 86177

Clinical Protocol BMS-986177 CV010010 FXIa

| SUMMARY OF K | EY CHANGES FOR REVISE |
|---|---|
| Section Number<br>& Title | Description of Change |
| Assignment and<br>Section 7.3:<br>Blinding | |
| Section 7.7.1:<br>Prohibited and/or<br>Restricted<br>Treatments | Prohibited/restricted<br>treatments were updated. |
| Section 8.1:<br>Discontinuation<br>from Study<br>Treatment | Updated the discontinuation criteria on events of complete clotting of hemodialysis circuit to include enoxaparin treatment arm and 5 or more patients. |
| Section 9.5:<br>Pharmacokinetics | Updates to further clarify<br>Table 9.5-1 were made. |
| Section 9.6:<br>Pharmacodynami<br>cs | Updates to further clarify<br>Table 9.6-1 and Table 9.6-2<br>were made. |
| Section 9.8:<br>Biomarker | Updates to further clarify Table 9.8-1 and Table 9.8-2 were made. Also, to remove clotting assessment from the blood line and URR. Kt/V assessment was further clarified. |
| All | Minor formatting and typographical corrections. One additional reference was added. Additional abbreviations were added to Appendix 1. |

Clinical Protocol CV010010
BMS-986177 FXIa

#### STUDY ACKNOWLEDGMENT/DISCLOSURE

I understand that this protocol contains information that is confidential and proprietary to Bristol-Myers Squibb Company (BMS). Any supplemental information that may be added to this document is also confidential and proprietary to BMS and must be kept in confidence in the same manner as the contents of this protocol.

I have read the original protocol/revised protocol and agree that it contains all necessary details for carrying out the study as described. I will conduct this protocol as outlined therein and will make a reasonable effort to complete the study within the time designated.

I will provide copies of the protocol and access to all information furnished by BMS to study personnel under my supervision. I will discuss this material with them to ensure that they are fully informed about the investigational product and the study.

I will provide protocol information to my Institutional Review Board(s) [IRB(s)] or Independent Ethics Committee(s) [IEC(s], I understand that original protocol/revised protocols must be reviewed by the Institutional Review Board or Independent Ethics Committee overseeing the conduct of the study and approved or given favorable opinion by all necessary Health Authorities before implementation unless to eliminate an immediate hazard to subjects.

I agree that the contents of the protocol may not be disclosed to any other person or entity or used for any other purpose without the prior written consent of BMS. The foregoing shall not apply to disclosure required by governmental regulations or laws; however, I will give prompt notice to BMS of any such disclosure.

I agree that the study data derived from this protocol may only be used and disclosed in furtherance of the protocol, for the medical treatment of a study subject or for publication of study results in accordance with the terms of the CTAg or as otherwise permitted by the terms of the CTAg.

I agree not to collect or use samples (e.g., tissue, blood, serum, urine) or collect data (other than for diagnostic or treatment purposes) from the study subjects while enrolled in the study, except as expressly permitted by the protocol or the terms of the CTAg.

I understand that I may terminate or suspend enrollment of the study at any time if it becomes necessary to protect the best interests of the study subjects. Unless otherwise provided in the CTAg, the study may be terminated at any time by BMS, with or without cause.

| Original Protocol | Revised Protocol |
|---|---|
| Protocol Number: CV010010 Site Number: 0003 | |
| Date of Protocol: September 06, 2017 | |
| ND Number: 130,436 EUDRACT Number: | NA |
| (signature) Jolene Kay Berg, MD (printed name*) | Date <u>215EP</u> <b>1</b> 017 |


This document contains information confidential and proprietary to Bristol-Myers Squibb

1